CLINICAL TRIAL: NCT03656510
Title: A Phase 2, Double-blind, Placebo-controlled Study to Evaluate the Antiviral Activity, Clinical Outcomes, Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Relationships of Different Doses of JNJ-53718678 in Children >=28 Days and <=3 Years of Age With Acute Respiratory Tract Infection Due to Respiratory Syncytial Virus Infection
Brief Title: Study to Evaluate Safety and Antiviral Activity of Doses of JNJ-53718678 in Children (>=28 Days to <=3 Years) With Respiratory Syncytial Virus Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Janssen made the strategic decision to discontinue the CROCuS study. This decision is not based on any safety concerns.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108520; 2016-003642-93 (EudraCT Number); 53718678RSV2002 (Other: Janssen Research & Development, LLC)
Expanded Access: NCT04221412 (No longer available)
Record Dates: First submitted 2018-08-15; First posted 2018-09-04 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — JNJ-53718678

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose: JNJ-53718678 (Experimental): Participants will be randomized to receive JNJ-53718678 2.5 milligram per kilogram (mg/kg) (Age Group 1: greater than or equal to [>=] 28 days and less than [<] 3 months of age), 3 mg/kg (Age Group 2: >=3 months and <6 months of age) and 4.5 mg/kg (Age Group 3: >=6 months and less than or equal to [<=3] years of age) orally twice daily for 7 days.
  Interventions: Drug: JNJ-53718678
- Low Dose: JNJ-53718678 (Experimental): Participants will be randomized to receive JNJ-53718678 0.85 mg/kg (Age Group 1: >=28 days and <3 months of age), 1 mg/kg (Age Group 2: >=3 months and <6 months of age) and 1.5 mg/kg (Age Group 3: >=6 months and 3 years of age) orally twice daily for 7 days.
  Interventions: Drug: JNJ-53718678
- Placebo (Placebo Comparator): Participants will be randomized to receive matching placebo (i.e. high volume placebo or low volume placebo to match the calculated volume of the JNJ-53718678 for the high dose or low dose) orally twice daily for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-53718678 — Participants will receive JNJ-53718678 (high dose or low dose) orally twice daily for 7 days.
  Arms: High Dose: JNJ-53718678; Low Dose: JNJ-53718678
Drug: Placebo — Participants will receive matching placebo (high volume or low volume) orally twice daily for 7 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the antiviral activity, clinical outcomes, safety, tolerability, and pharmacokinetic/pharmacodynamic relationships of different oral dose levels of JNJ-53718678 in children greater than or equal to 28 days and less than or equal to 3 years of age with respiratory syncytial virus (RSV) disease (hospitalized participants [Cohort 1] or outpatients [Cohort 2]).

DETAILED DESCRIPTION:
JNJ-53718678 is an investigational respiratory syncytial virus (RSV) specific fusion inhibitor and is under development for the treatment of RSV infection, which results in an upper and/or lower respiratory tract illness. The primary hypothesis of this study is that JNJ-53718678 has antiviral activity against RSV (that is, results in a decrease in RSV nasal viral load from immediately prior to first dose of study drug until Day 5). This will be assessed by a positive dose-response relationship of JNJ-53718678 compared to placebo. Besides the RSV nasal viral load through day 5, other timepoints will also be evaluated as well as other nasal viral load related parameters. In addition, the evolution of signs and symptoms of RSV disease will be evaluated. Participants' safety will be monitored throughout the study by evaluating the occurrence and severity of adverse events and by laboratory and electrocardiogram measurements. Study participants will be identified when they are hospitalized or expected to be hospitalized within 24 hours after presentation to the hospital (Cohort 1) or present for medical care as outpatients (Cohort 2) with symptoms of an acute respiratory illness supporting a diagnosis of RSV infection. Eligible participants will be randomized 1:1:1 to receive either a low or a high dose of JNJ 53718678 or placebo and will be receiving study treatment for 7 days. They will be followed up for 3 weeks after the last dose. The total study duration for each participant will be approximately 29 days.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form (ICF) must be given
* Laboratory diagnosis of respiratory syncytial virus (RSV) infection
* The participant has an acute respiratory illness
* The time of onset of RSV symptoms to the anticipated time of randomization must be less than or equal to (<=) 5 days
* Except for the RSV-related illness, the Participant must be medically stable in case of allowed co-morbid conditions
* The participant must have been assessed per local public health practice and considered not to have Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection during this respiratory infection

Exclusion Criteria:

* The participant is less than (<) 3 months postnatal age at screening and was born prematurely (i.e, <37 weeks and 0 days of gestation) OR if the participant weighs <2.4 kilogram (kg) or greater than (>) 16.8 kg
* Participant is considered by the investigator to be immunocompromised within the past 12 months
* Participant unwilling or unable to undergo mid-turbinate nasal swab procedures
* Participant is receiving chronic home oxygen therapy at screening
* Participant has other clinically significant abnormal electrocardiogram (ECG) findings not consistent with the present risk factor for severe RSV disease (if applicable) in the study population, as judged by the investigator based on the machine read ECG results at screening
* The participant has a QTcF interval greater than (>)450 millisecond (ms) per the machine read (mean of triplicate) parameter result confirmed by repeat triplicate ECG recording during screening

Ages: 28 Days to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 246 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (169):
- United States (14):
  - Madera Family Medical Group, Madera, California
  - FOMAT Medical Research, Ventura, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Elite Clinical Trials, Blackfoot, Idaho
  - Saltzer Medical Group, Nampa, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Craig A. Spiegel, MD, Bridgeton, Missouri
  - SUNY Upstate Medical University - Upstate Golisano Children's Hospital (GCH), Syracuse, New York
  - Santiago Reyes, MD, Oklahoma City, Oklahoma
  - Coastal Pediatric Research, Summerville, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
  - West Virginia University, Morgantown, West Virginia
- Argentina (9):
  - Hospital Italiano Regional Del Sur, Bahía Blanca
  - Fundación Respirar, Buenos Aires
  - Hospital Central Militar Cirujano Mayor Dr Cosme Argerich, Buenos Aires
  - CEMIC (Centro de Educación Médica e Investigaciones Clínicas), City of Buenos Aires
  - Hospital Pedro de Elizalde, City of Buenos Aires
  - Hospital Italiano de La Plata, Ciudad de La Plata
  - Hospital Universitario Austral, Pilar
  - Hospital del Niño Jesús, San Miguel de Tucumán
  - Clinica Mayo de UMCB, San Miguel de Tucumán
- Belgium (3):
  - ULB Hôpital Erasme, Anderlecht
  - UZ Antwerpen, Edegem
  - C.H.R. Citadelle, Liège
- Brazil (13):
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Fundacao para o Desenvolvimento Medico Hospitalar (UNESP Botucatu), Botucatu
  - Sociedade Campineira de Educacao e Instrucao Hospital e Maternidade Celso Pierro, Campinas
  - Nucleo de Pesquisa do Hospital Pequeno Princípe, Curitiba
  - Secretaria da Saude do Estado do Ceara - Hospital Doutor Carlos Alberto Studart Gomes, Fortaleza
  - Centro de Estudos e Pesquisas em Moléstias Infecciosas - CEPCLIN, Natal
  - Associacao Hospitalar Beneficente Sao Vicente de Paulo - Hospital Sao Vicente de Paulo, Passo Fundo
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Fundacao Jose Luiz Egydio Setubal, São Paulo
  - CMPC - Consultoria Médica e Pesquisa Clínica, Sorocaba
  - Santa Casa de Misericórdia de Votuporanga, Votuporanga
- Bulgaria (8):
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - UMHAT 'Sveti Georgi'-Plovdiv, Plovdiv
  - UMHAT 'Kanev' EAD, Rousse
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - DCC 'Sv. Vrach and Sv. Sv. Kuzma and Damyan', OOD, Sofia
  - UMHAT 'Aleksandrovska' EAD, Sofia
  - SHATCD 'Prof. Ivan Mitev' EAD, Sofia
- France (7):
  - CHU de Caen, Caen
  - Hopital Antoine Beclere, Clamart
  - CHU de Montpellier - Arnaud de Villeneuve, Montpellier
  - CHU de Nantes hotel Dieu, Nantes
  - Hopitaux pediatriques CHU Lenval, Nice
  - Hôpital Necker-Enfants Malades, Paris
  - Hopital Charles Nicolle, Rouen
- Germany (5):
  - Kinderarztpraxis Bramsche, Bramsche
  - Hürthpark Kinder & Jugendärzte, Hürth
  - Praxiszentrum Triftplatz, Schönau am Königssee
  - Kinderärztliche Gemeinschaftspraxis, Wolfsburg
  - Universitatsklinikum Wurzburg, Würzburg
- Hungary (9):
  - Semmelweis Egyetem, II. sz. Gyermekgyógyászati Klinika, Budapest
  - Del Pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet Szent Laszlo Telephely, Budapest
  - Debreceni Egyetem Klinikai Központ,Infektológiai Klinika, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Futurenest Klinikai Kutato Kft., Miskolc
  - Kanizsai Dorottya Kórház, Nagykanizsa
  - Szegedi Tudomanyegyetem, Szeged
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktatokorhaz, Székesfehérvár
  - Csolnoky Ferenc Korhaz, Veszprém
- Italy (7):
  - A O U Sant Orsola Malpighi, Bologna
  - Università degli Studi di Milano, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - ASST Fatebenefratelli Sacco / Ospedale dei Bambini V. Buzzi, Milan
  - Dipartimento di Pediatria dell'Ospedale Luigi Sacco, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Department of Pediatrics University of Pavia, Policlinico San Matteo, Pavia
  - Ospedale degli Infermi, Ponderano
- Japan (19):
  - Hosaka Kodomo Clinic, Bunkyō City
  - Kobayashi Pediatric Clinic, Fujieda
  - Fukui-ken Saiseikai Hospital, Fukui
  - National Hospital Organization Fukuyama Medical Center, Fukuyama
  - Fukuyama City Hospital, Fukuyama
  - Tanabe Pediatrics Clinic, Hatsukaichi
  - Kagoshima Children's Hospital, Hioki
  - National Hospital Organization Hirosaki General Medical Center, Hirosaki
  - Shirao Clinic of Pediatrics and Pediatric Allergy, Hiroshima
  - National Hospital Organization Kanazawa Medical Center, Kanazawa
  - Kojunkai Daido Clinic, Nagoya
  - Kojunkai Daido Hospital, Nagoya
  - Momotaro Clinic, Okayama
  - National Hospital Organization Beppu Medical Center, Ōita
  - National Hospital Organization Saitama National Hospital, Saitama
  - KKR Sapporo Medical Center, Sapporo
  - Tsuda Pediatrics Clinic, Setagaya-ku
  - Okawa Children & Family Clinic, Tokyo
  - INAMI Pediatric clinic, Tokyo
- Malaysia (4):
  - Hospital Selayang, Batu Caves
  - Hospital Miri, Miri
  - Hospital Tuanku Fauziah, Pusat Bandar Kangar
  - Hospital Sibu, Sibu
- Mexico (5):
  - RM Pharma Specialists, Benito Juárez
  - Instituto Nacional de Pediatría, Coyoacán
  - Hospital Civil de Guadalajara, Guadalajara
  - Hospital Infantil de Mexico Federico Gomez, Mexico City
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
- Poland (7):
  - Osrodek Badan Klinicznych In-Vivo Sp. z o.o., Bydgoszcz
  - Zespol Opieki Zdrowotnej w Debicy, Oddzial Dzieciecy, Dębica
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Oddzial Pediatrii i Neurologii Dzieciecej, Krakow
  - Instytut Gruzlicy i Chorob Pluc Oddzial Terenowy im. Rudnikow w Rabce-Zdroj, Oddzial Pulmonologii, Rabka-Zdrój
  - ALERGO-MED Specjalistyczna Przychodnia Lekarska Sp. z o.o., Tarnów
  - Szpital im Swietej Jadwigi Slaskiej Oddzial Pediatryczny z Pododdzialem Niemowlecym, Trzebnica
  - NZOZ Salmed, Łęczna
- Russia (11):
  - Infectious Clinical Hospital #1 Of The Moscow City Health Department, Moscow
  - OOO MDP-Medical Group, Odintsovo
  - City Children Clinical Outpatient Clinic #5, Perm
  - OOO 'Medical Technologies', Saint Petersburg
  - Children Outpatient Clinic 45 Of Nevskiy Region, Saint Petersburg
  - OOO 'Arsvite North-West', Saint Petersburg
  - LLC Pitercliniсa, Saint Petersburg
  - LLC Kurator, Saint Petersburg
  - Siberian State Medical University, Tomsk
  - Bashkir State Medical University, Ufa
  - Yaroslavl State Medical University Based On Children Polyclinics #5, Yaroslavl
- South Africa (4):
  - Tygrberg Hospital, Bellville
  - Josha Research, Bloemfontein
  - VX Pharma, Pretoria
  - Two Military Hospital, Wynberg
- South Korea (4):
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
- Spain (13):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Del Mar, Barcelona
  - Hosp. Univ. de Burgos, Burgos
  - Hosp. Univ. de Getafe, Getafe
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Puerta Del Sur, Móstoles
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
- Sweden (3):
  - Barn- Och Ungdomsmedicin, Malmo
  - Sachsska barn-och ungdomssjukhuset, Stockholm
  - Astrid Lindgrens barnsjukhus Solna, Stockholm
- Taiwan (6):
  - Hsinchu MacKay Memorial Hospital, Hsinchu
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Chang Gung Memorial Hospital- Linkou, Taoyuan
- Thailand (6):
  - Queen Sirikit National Institute of Child Health, Bangkok
  - Tropical Medicine Hospital, Mahidol University, Bangkok
  - Siriraj Hospital Mahidol University, Bangkok
  - Chiang Mai University, Chiang Mai
  - Research Institute for Health Sciences, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
- Turkey (Türkiye) (9):
  - Cukurova University Medical Faculty Balcali Hospital, Adana
  - Ankara University Medical Faculty, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Gazi University Medical Faculty, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Ege University Medical Faculty, Izmir
  - Saglik Bilimleri University Sariyer Hamidiye Etfal Training and Research Hospital, Sarıyer
  - Karadeniz Teknik University Medical Faculty, Trabzon
- United Kingdom (3):
  - Royal Devon & Exeter Hospital, Exeter
  - Whipps Cross University Hospital, London
  - The Adam Practice, Poole

REFERENCES:
- [Derived] Ferrero F, Lin CY, Liese J, Luz K, Stoeva T, Nemeth A, Gijon M, Calvo C, Natalini S, Toh TH, Deleu S, Chen B, Rusch S, Sanchez BL, Leipoldt I, Vijgen L, Huntjens D, Baguet T, Bertzos K, Gamil M, Stevens M; CROCuS Investigators. CROCuS, a Phase II Study Evaluating the Antiviral Activity, Clinical Outcomes, and Safety of Rilematovir in Children Aged >/= 28 Days and </= 3 Years with Acute Respiratory Tract Infection Due to Respiratory Syncytial Virus. Paediatr Drugs. 2024 Jul;26(4):411-427. doi: 10.1007/s40272-024-00625-x. Epub 2024 Apr 22. PMID 38649595

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Placebo: Participants of age groups (age group 1: greater than or equal to [>=] 28 days to less than [<] 3 months, age group 2: >=3 months to <6 months, and age group 3: >=6 months to less than or equal to [<=] 3 years), who were hospitalized or expected to be hospitalized within 24 hours after presentation to the hospital received placebo matching to JNJ-53718678 (high volume placebo or low volume placebo to match the calculated volume of the JNJ-53718678 for the high dose or low dose, respectively) orally once daily for 7 days.
- Cohort 1: JNJ-53718678 Low Dose: Participants who were hospitalized or expected to be hospitalized within 24 hours after presentation to the hospital received JNJ-53718678 1.7 milligrams per kilogram (mg/kg) for age group 1: >=28 days to <3 months; 2 mg/kg for age group 2: >=3 months to <6 months; and 3 mg/kg for age group 3: >=6 months to <=3 years, orally once daily for 7 days.
- Cohort 1: JNJ-53718678 High Dose: Participants who were hospitalized or expected to be hospitalized within 24 hours after presentation to the hospital received JNJ-53718678 5 mg/kg for age group 1: >=28 days to <3 months; 6 mg/kg for age group 2: >=3 months to <6 months; and 9 mg/kg for age group 3: >=6 months to <=3 years, orally once daily for 7 days.
- Cohort 2: Placebo: As per the original dosing, outpatients of age groups (age group 1: >=28 days to <3 months, age group 2: >=3 months to <6 months, and age group 3: >=6 months to <=3 years) were randomized to receive placebo matching to JNJ-53718678 (high volume placebo or low volume placebo to match the calculated volume of the JNJ-53718678 for the high dose or low dose, respectively) orally once daily for 7 days. After protocol amendment 4, participants received placebo matching to JNJ-53718678 (high dose or low dose) orally twice daily for 7 days.
- Cohort 2: JNJ-53718678 Low Dose: As per the original dosing, outpatients were randomized to receive JNJ-53718678 1.7 mg/kg for age group 1: >=28 days to <3 months; 2 mg/kg for age group 2: >=3 months to <6 months; and 3 mg/kg for age group 3: >=6 months to <=3 years, orally once daily for 7 days. After protocol amendment 4, participants were randomized to receive JNJ-53718678 0.85 mg/kg for age group 1, JNJ-53718678 1.0 mg/kg for age group 2, and JNJ-53718678 1.5 mg/kg for age group 3, orally twice daily for 7 days.
- Cohort 2: JNJ-53718678 High Dose: As per the original dosing, outpatients were randomized to receive JNJ-53718678 5 mg/kg for age group 1: >=28 days to <3 months; 6 mg/kg for age group 2: >=3 months to <6 months; and 9 mg/kg for age group 3: >=6 months to <=3 years, orally once daily for 7 days. After protocol amendment 4, participants were randomized to receive JNJ-53718678 2.5 mg/kg for age group 1, JNJ-53718678 3.0 mg/kg for age group 2, and JNJ-53718678 4.5 mg/kg for age group 3, orally twice daily for 7 days.
Period: Overall Study
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Started | 50 | 49 | 48 | 34 | 34 | 31
Completed | 48 | 48 | 48 | 33 | 34 | 31
Not Completed | 2 | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose | Total
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31 | 246
Age, Continuous [Mean (Standard Deviation); unit: months] | 8.4 (8.59) | 8.6 (8.74) | 8.5 (8.21) | 13.8 (10.31) | 14.8 (10.9) | 17.2 (8.81) | 11.2 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 23 | 13 | 8 | 14 | 101
  Male | 27 | 29 | 25 | 21 | 26 | 17 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 19 | 21 | 10 | 9 | 10 | 87
  Not Hispanic or Latino | 29 | 28 | 24 | 24 | 25 | 21 | 151
  Unknown or Not Reported | 3 | 2 | 3 | 0 | 0 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 1 | 0 | 0 | 0 | 5
  Asian | 15 | 14 | 11 | 11 | 14 | 13 | 78
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 0 | 1 | 0 | 0 | 5
  White | 28 | 29 | 31 | 22 | 19 | 18 | 147
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 4 | 1 | 4 | 0 | 1 | 0 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 5 | 5 | 6 | 0 | 0 | 0 | 16
  BRAZIL | 1 | 5 | 3 | 7 | 5 | 5 | 26
  BULGARIA | 3 | 0 | 2 | 6 | 6 | 7 | 24
  GERMANY | 0 | 1 | 2 | 0 | 0 | 0 | 3
  HUNGARY | 2 | 2 | 4 | 3 | 2 | 0 | 13
  ITALY | 1 | 1 | 1 | 0 | 0 | 0 | 3
  JAPAN | 5 | 3 | 4 | 8 | 12 | 7 | 39
  MALAYSIA | 4 | 2 | 4 | 1 | 0 | 1 | 12
  MEXICO | 0 | 0 | 0 | 0 | 1 | 2 | 3
  POLAND | 0 | 0 | 0 | 1 | 1 | 0 | 2
  RUSSIAN FEDERATION | 1 | 1 | 0 | 0 | 0 | 0 | 2
  SOUTH AFRICA | 0 | 0 | 0 | 1 | 0 | 0 | 1
  SOUTH KOREA | 2 | 0 | 0 | 0 | 0 | 0 | 2
  SPAIN | 17 | 17 | 20 | 5 | 3 | 3 | 65
  SWEDEN | 2 | 1 | 0 | 0 | 0 | 0 | 3
  TAIWAN | 3 | 5 | 2 | 0 | 0 | 2 | 12
  THAILAND | 1 | 3 | 0 | 2 | 2 | 2 | 10
  TURKEY | 3 | 1 | 0 | 0 | 0 | 0 | 4
  UNITED KINGDOM | 0 | 2 | 0 | 0 | 0 | 0 | 2
  UNITED STATES | 0 | 0 | 0 | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Syncytial Virus (RSV) Viral Load Area Under Curve (AUC) From Immediately Prior to First Dose of Study Drug (Baseline) Through Day 5 (AUC[Day 5])
Description: RSV viral load AUC from immediately prior to first dose of study drug through Day 5 was determined. The RSV viral load was measured by quantitative reverse transcription polymerase chain reaction (qRT-PCR) assay in mid-turbinate nasal swab specimens. As planned, combined data for both the cohorts was collected, analyzed and reported for this outcome measure.
Time Frame: Baseline through Day 5
Population: Intent-to-Treat-infected (ITT-i) analysis set included all randomized participants who received at least one dose of study drug and who had a centrally confirmed RSV RNA viral load of greater than or equal to (>=) 1 log10 copies/mL above the lower limit of quantification (LLOQ) of the RSV RT-qPCR assay at baseline. Analyses on the ITT-i set were performed as randomized.
Measure: Mean (95% Confidence Interval); unit: log10 copies*day per milliliter (mL)
Groups:
- Cohorts 1 and 2: Placebo: As per the original dosing, participants of age groups (age group 1: >=28 days to <3 months, age group 2: >=3 months to <6 months, and age group 3: >=6 months to less than or equal to [<=3] years) were randomized to receive placebo matching to JNJ-53718678 (high volume placebo or low volume placebo to match the calculated volume of the JNJ-53718678 for the high dose or low dose, respectively) orally once daily for 7 days in Cohorts 1 and 2. After protocol amendment 4, participants in Cohort 2 were randomized to receive placebo matching to JNJ-53718678 (high dose or low dose) orally twice daily for 7 days.
- Cohorts 1 and 2: JNJ-53718678 Low Dose: As per the original dosing, participants were randomized to receive JNJ-53718678 1.7 mg/kg for age group 1: >=28 days to <3 months; 2 mg/kg for age group 2: >=3 months to <6 months; and 3 mg/kg for age group 3: >=6 months to <=3 years, orally once daily for 7 days in Cohorts 1 and 2. After protocol amendment 4, participants in Cohort 2 were randomized to receive JNJ-53718678 0.85 mg/kg for age group 1, JNJ-53718678 1.0 mg/kg for age group 2, and JNJ-53718678 1.5 mg/kg for age group 3, orally twice daily for 7 days.
- Cohorts 1 and 2: JNJ-53718678 High Dose: As per the original dosing, participants were randomized to receive JNJ-53718678 5 mg/kg for age group 1: >=28 days to <3 months; 6 mg/kg for age group 2: >=3 months to <6 months; and 9 mg/kg for age group 3: >=6 months to <=3 years, orally once daily for 7 days in Cohorts 1 and 2 . After protocol amendment 4, participants in Cohort 2 were randomized to receive JNJ-53718678 2.5 mg/kg for age group 1, JNJ-53718678 3.0 mg/kg for age group 2, and JNJ-53718678 4.5 mg/kg for age group 3, orally twice daily for 7 days.
Arm/Group | Cohorts 1 and 2: Placebo | Cohorts 1 and 2: JNJ-53718678 Low Dose | Cohorts 1 and 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 79 | 80 | 72
log10 copies*day per milliliter (mL) | 22.74 [21.677 to 23.800] | 21.48 [20.402 to 22.566] | 21.51 [20.374 to 22.650]

2. Secondary Outcome: RSV Viral Load Over Time
Description: RSV viral load actual values over time were measured by qRT-PCR in the nasal swab specimens collected at the clinic visits and at home. As planned, combined data for both the cohorts was collected, analyzed and reported for this outcome measure.
Time Frame: Baseline, Days 3, 5, 8, 14, and 21
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had centrally confirmed RSV RNA viral load of >=1 log10 copies/mL above the LLOQ of the RSV RT-qPCR assay at baseline. Analyses on ITT-i set were performed as randomized. Here, 'n' (number analyzed) represents number of participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Cohorts 1 and 2: Placebo | Cohorts 1 and 2: JNJ-53718678 Low Dose | Cohorts 1 and 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 79 | 80 | 72
log10 copies/mL
  Baseline | 6.913 (1.3449) | 7.113 (1.3667) | 7.004 (1.4709)
  Day 3: number analyzed (Participants) | 77 | 79 | 71
  Day 3 | 5.398 (1.5834) | 5.432 (1.8952) | 5.271 (1.7710)
  Day 5: number analyzed (Participants) | 77 | 77 | 72
  Day 5 | 4.146 (1.8508) | 4.079 (1.8760) | 3.883 (1.9815)
  Day 8: number analyzed (Participants) | 78 | 73 | 70
  Day 8 | 2.604 (2.0857) | 2.108 (1.8538) | 2.078 (1.8319)
  Day 14: number analyzed (Participants) | 73 | 74 | 67
  Day 14 | 1.640 (1.9515) | 1.636 (2.2221) | 1.440 (1.8768)
  Day 21: number analyzed (Participants) | 74 | 78 | 68
  Day 21 | 1.150 (1.7752) | 0.817 (1.5347) | 0.810 (1.6699)

3. Secondary Outcome: Change From Baseline in RSV Viral Load Over Time
Description: Change from baseline in RSV viral load over time was measured by qRT-PCR in the nasal swab specimens collected at the clinic visits and at home. As planned, combined data for both the cohorts was collected, analyzed and reported for this outcome measure.
Time Frame: Baseline up to Days 3, 5, 8, 14, and 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Cohorts 1 and 2: Placebo | Cohorts 1 and 2: JNJ-53718678 Low Dose | Cohorts 1 and 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 79 | 80 | 72
log10 copies/mL
  Day 3: number analyzed (Participants) | 77 | 79 | 71
  Day 3 | -1.502 (1.3290) | -1.690 (1.6225) | -1.694 (1.5134)
  Day 5: number analyzed (Participants) | 77 | 77 | 72
  Day 5 | -2.754 (1.7699) | -3.049 (1.6493) | -3.121 (1.8453)
  Day 8: number analyzed (Participants) | 78 | 73 | 70
  Day 8 | -4.308 (2.2435) | -5.017 (1.8563) | -4.948 (1.8428)
  Day 14: number analyzed (Participants) | 73 | 74 | 67
  Day 14 | -5.292 (2.2968) | -5.471 (2.4289) | -5.578 (2.2707)
  Day 21: number analyzed (Participants) | 74 | 78 | 68
  Day 21 | -5.801 (2.1652) | -6.302 (2.0439) | -6.268 (1.9394)

4. Secondary Outcome: Least Squares (LS) Mean RSV Viral Load on Days 3, 8 and 14
Description: LS mean RSV viral load on Days 3, 8, and 14 was reported. LS mean viral load (log10 copies/mL) was estimated per time point. The difference in RSV viral Load AUC (log10 copies*day/mL) from immediately prior to first dose of study drug (baseline) through Day 3, 8 and 14 was determined from the model estimating the LS Mean Viral Load per time point, and is presented in the statistical analysis. The RSV viral load was measured by qRT-PCR assay in mid-turbinate nasal swab specimens. As planned, combined data for both the cohorts was collected, and analyzed for this outcome measure at Days 3 and 8, however combined Cohort 1 and Cohort 2 data were not analyzed for this outcome measure at Day 14, due to the premature study termination.
Time Frame: Baseline through Days 3, 8, and 14
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies*day/mL
Arm/Group | Cohorts 1 and 2: Placebo | Cohorts 1 and 2: JNJ-53718678 Low Dose | Cohorts 1 and 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 79 | 80 | 72
log10 copies*day/mL
  Day 3: LS means RSV Viral Load | 5.48 [5.129 to 5.834] | 5.36 [5.009 to 5.717] | 5.32 [4.949 to 5.695]
  Day 8: LS means RSV Viral Load | 2.66 [2.307 to 3.011] | 2.08 [1.716 to 2.444] | 2.08 [1.701 to 2.450]
  Day 14: LS means RSV Viral Load: number analyzed (Participants) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Cohorts 1 and 2: Placebo vs Cohorts 1 and 2: JNJ-53718678 Low Dose; Difference versus placebo in mean RSV viral load AUC on Day 3; Test type: Other; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-1.382 to 0.185]
Statistical Analysis 2: Comparison: Cohorts 1 and 2: Placebo vs Cohorts 1 and 2: JNJ-53718678 High Dose; Difference versus placebo in mean RSV viral load AUC on Day 3; Test type: Other; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.190 to 0.418]
Statistical Analysis 3: Comparison: Cohorts 1 and 2: Placebo vs Cohorts 1 and 2: JNJ-53718678 Low Dose; Difference versus placebo in mean RSV viral load AUC on Day 8; Test type: Other; Mean Difference (Final Values) = -2.46, 95% CI 2-sided [-4.674 to -0.250]
Statistical Analysis 4: Comparison: Cohorts 1 and 2: Placebo vs Cohorts 1 and 2: JNJ-53718678 High Dose; Difference versus placebo in mean RSV viral load AUC on Day 8; Test type: Other; Mean Difference (Final Values) = -2.38, 95% CI 2-sided [-4.645 to -0.114]

5. Secondary Outcome: Time to Undetectable RSV Viral Load
Description: Time to undetectable RSV viral load (as measured by qRT-PCR) was defined as the time in hours from first dose of study drug to first post-baseline timepoint at which the virus was undetectable and after which there were no more detectable virus assessments. As planned, combined data for both the cohorts was collected, analyzed and reported for this outcome measure.
Time Frame: Up to Day 21
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had centrally confirmed RSV RNA viral load of >=1 log10 copies/mL above the LLOQ of the RSV RT-qPCR assay at baseline. Analyses on ITT-i set were performed as randomized.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Cohorts 1 and 2: Placebo | Cohorts 1 and 2: JNJ-53718678 Low Dose | Cohorts 1 and 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 79 | 80 | 72
Hours | 467.0 [332.90 to 478.40] | 428.3 [309.50 to 480.40] | 330.7 [308.28 to 476.00]

6. Secondary Outcome: Percentage of Participants With Undetectable RSV Viral Load at Each Timepoint Throughout the Study
Description: Percentage of participants with undetectable RSV viral load (as measured by qRT-PCR) at each timepoint throughout the study was reported. As planned, combined data for both the cohorts were collected, analyzed and reported for this outcome measure.
Time Frame: Baseline, Days 3, 5, 8, 14 and 21
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Cohorts 1 and 2: Placebo | Cohorts 1 and 2: JNJ-53718678 Low Dose | Cohorts 1 and 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 79 | 80 | 72
Percentage of participants
  Baseline | 0 | 0 | 0
  Day 3: number analyzed (Participants) | 77 | 79 | 71
  Day 3 | 1.3 | 3.8 | 2.8
  Day 5: number analyzed (Participants) | 77 | 77 | 72
  Day 5 | 7.8 | 9.1 | 11.1
  Day 8: number analyzed (Participants) | 78 | 73 | 70
  Day 8 | 33.3 | 38.4 | 38.6
  Day 14: number analyzed (Participants) | 73 | 74 | 67
  Day 14 | 54.8 | 58.1 | 58.2
  Day 21: number analyzed (Participants) | 74 | 78 | 68
  Day 21 | 67.6 | 76.9 | 77.9

7. Secondary Outcome: Change From Baseline in Parent(s)/Caregiver(s) Pediatric RSV Electronic Severity and Outcomes Rating System (PRESORS) Scores
Description: PRESORS is a questionnaire recording presence and severity of signs and symptoms of RSV disease (fever, cough, sputum, wheezing, difficulty breathing, nasal congestion, and feeding issues). PRESORS overall RSV symptoms summary parameter consisted of 12-items, each item score ranges from 0 to 3. A summary score was derived (mean of the item scores) which also ranges from 0 to 3. The higher the score, the worse the symptom.
Time Frame: Baseline up to Days 3, 5, 8, 14 and 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44 | 32 | 33 | 28
Units on a scale
  Day 3: number analyzed (Participants) | 45 | 40 | 41 | 25 | 27 | 26
  Day 3 | -0.51 (0.571) | -0.55 (0.618) | -0.70 (0.594) | -0.25 (0.576) | -0.15 (0.427) | -0.21 (0.537)
  Day 5: number analyzed (Participants) | 45 | 41 | 41 | 28 | 27 | 26
  Day 5 | -0.91 (0.585) | -0.88 (0.542) | -1.11 (0.581) | -0.48 (0.572) | -0.52 (0.558) | -0.58 (0.644)
  Day 8: number analyzed (Participants) | 44 | 41 | 41 | 28 | 27 | 26
  Day 8 | -1.15 (0.581) | -1.25 (0.537) | -1.39 (0.514) | -0.85 (0.526) | -0.83 (0.582) | -1.04 (0.628)
  Day 14: number analyzed (Participants) | 44 | 39 | 40 | 28 | 27 | 26
  Day 14 | -1.40 (0.591) | -1.39 (0.582) | -1.59 (0.458) | -1.06 (0.529) | -1.08 (0.568) | -1.24 (0.681)
  Day 21: number analyzed (Participants) | 42 | 40 | 41 | 28 | 26 | 26
  Day 21 | -1.41 (0.637) | -1.33 (0.559) | -1.56 (0.468) | -1.12 (0.529) | -1.15 (0.496) | -1.29 (0.596)

8. Secondary Outcome: Change From Baseline in Clinician PRESORS Score
Description: Change from baseline in clinician PRESORS scores (for concepts: activity level, sleep disturbance, breathing problems, retractions, tachypnea, feeding problem, cough, nasal secretions, wheezing, dehydration) was assessed. Clinician PRESORS is a questionnaire recording presence and severity of signs and symptoms of RSV disease and consisted of 10-items, each item score ranges from 0 to 3. Overall RSV symptoms summary parameter was derived (mean of the item scores) which also ranges from 0 to 3. The higher the score, the worse the symptom.
Time Frame: Baseline, up to Days 3, 5, 8, 14 and 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44 | 32 | 33 | 28
Units on a scale
  Day 3: number analyzed (Participants) | 43 | 41 | 42 | 29 | 29 | 26
  Day 3 | -0.45 (0.441) | -0.45 (0.517) | -0.48 (0.469) | -0.25 (0.424) | -0.21 (0.378) | -0.29 (0.338)
  Day 5: number analyzed (Participants) | 42 | 38 | 41 | 28 | 28 | 25
  Day 5 | -0.73 (0.582) | -0.71 (0.424) | -0.83 (0.483) | -0.38 (0.415) | -0.37 (0.462) | -0.60 (0.516)
  Day 8: number analyzed (Participants) | 41 | 38 | 38 | 30 | 29 | 26
  Day 8 | -0.92 (0.461) | -1.04 (0.396) | -1.04 (0.449) | -0.71 (0.529) | -0.63 (0.423) | -0.85 (0.552)
  Day 14: number analyzed (Participants) | 40 | 37 | 34 | 28 | 27 | 23
  Day 14 | -1.10 (0.466) | -1.11 (0.428) | -1.14 (0.369) | -0.81 (0.497) | -0.77 (0.436) | -0.91 (0.541)
  Day 21: number analyzed (Participants) | 35 | 40 | 33 | 29 | 28 | 27
  Day 21 | -1.13 (0.424) | -1.12 (0.433) | -1.17 (0.336) | -0.87 (0.455) | -0.81 (0.411) | -0.93 (0.524)

9. Secondary Outcome: Time to Resolution of RSV Symptoms Based on PRESORS Caregiver (ObsRO)
Description: Time to resolution is defined as time from first dose of study drug until the first time of resolution of all RSV symptoms (breathing problems, retractions, tachypnea, breathing sounds, cough, tachycardia, nasal secretions, sleep disturbance, crying, illness behavior, feeding problems, and dehydration). Resolution occurs when all symptoms from the caregiver reported outcomes (ObsRO) are scored as none or mild (score of 0 or 1, respectively) for at least 24 hours.
Time Frame: Up to Day 21
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44 | 32 | 33 | 28
Hours | 193.5 [161.80 to 243.80] | 163.6 [108.70 to 198.70] | 151.8 [114.70 to 223.70] | 166.6 [141.50 to 207.20] | 206.1 [159.20 to 232.80] | 176.9 [148.30 to 264.20]

10. Secondary Outcome: Time to Improvement on Overall Health
Description: Time to improvement based on general questions on overall health was assessed. Time from first dose of study drug until first time status of improvement of RSV symptoms reported as "very much improved" or "much improved" based on response to question 'Would you say the child's RSV symptoms have improved, are about the same or are worse than when the child entered the study'.
Time Frame: Up to Day 21
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had centrally confirmed RSV RNA viral load of >=1 log10 copies/mL above the LLOQ of the RSV RT-qPCR assay at baseline. Analyses on ITT-i set were performed as randomized. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 45 | 44 | 43 | 32 | 32 | 28
Hours | 189.6 [187.80 to 192.50] | 190.2 [188.70 to 200.00] | 189.1 [186.90 to 191.90] | 186.8 [184.30 to 190.40] | 198.2 [185.30 to 237.30] | 187.9 [185.90 to 189.80]

11. Secondary Outcome: Percentage of Participants by Status of RSV Symptoms Based on PRESORS Caregiver (ObsRO) General Question Over Time
Description: Percentage of participants by status of RSV symptoms based on PRESORS caregiver (ObsRO) general question over time was assessed. PRESORS is a questionnaire recording presence and severity of signs and symptoms of RSV disease (fever, cough, sputum, wheezing, difficulty breathing, nasal congestion, and feeding issues). Status of RSV symptoms was assessed by a question (how would you rate the child's RSV symptoms now?) of PRESORS questionnaire and responses were categorized as: 1) none, 2) very mild, 3) mild, 4) moderate, 5) severe, and 6) very severe.
Time Frame: Baseline, Days 3, 5, 8, 14, and 21
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had centrally confirmed RSV RNA viral load of >=1 log10 copies/mL above LLOQ of RSV RT-qPCR assay at baseline. Analyses on ITT-i set were performed as randomized. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represents number of participants who were evaluable at specified timepoints.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44 | 32 | 33 | 28
Percentage of participants
  Baseline: None: number analyzed (Participants) | 45 | 43 | 41 | 28 | 27 | 26
  Baseline: None | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: Very mild: number analyzed (Participants) | 45 | 43 | 41 | 28 | 27 | 26
  Baseline: Very mild | 0 | 0 | 2.4 | 7.1 | 7.4 | 3.8
  Baseline: Mild: number analyzed (Participants) | 45 | 43 | 41 | 28 | 27 | 26
  Baseline: Mild | 6.7 | 7.0 | 4.9 | 32.1 | 22.2 | 19.2
  Baseline: Moderate: number analyzed (Participants) | 45 | 43 | 41 | 28 | 27 | 26
  Baseline: Moderate | 51.1 | 55.8 | 51.2 | 53.6 | 55.6 | 46.2
  Baseline: Severe: number analyzed (Participants) | 45 | 43 | 41 | 28 | 27 | 26
  Baseline: Severe | 37.8 | 27.9 | 41.5 | 7.1 | 14.8 | 30.8
  Baseline: Very severe: number analyzed (Participants) | 45 | 43 | 41 | 28 | 27 | 26
  Baseline: Very severe | 4.4 | 9.3 | 0 | 0 | 0 | 0
  Day 3: None: number analyzed (Participants) | 47 | 43 | 44 | 29 | 31 | 28
  Day 3: None | 0 | 2.3 | 0 | 3.4 | 0 | 0
  Day 3: Very mild: number analyzed (Participants) | 47 | 43 | 44 | 29 | 31 | 28
  Day 3: Very mild | 6.4 | 9.3 | 6.8 | 0 | 3.2 | 0
  Day 3: Mild: number analyzed (Participants) | 47 | 43 | 44 | 29 | 31 | 28
  Day 3: Mild | 23.4 | 18.6 | 36.4 | 27.6 | 19.4 | 25.0
  Day 3: Moderate: number analyzed (Participants) | 47 | 43 | 44 | 29 | 31 | 28
  Day 3: Moderate | 46.8 | 48.8 | 43.2 | 62.1 | 64.5 | 64.3
  Day 3: Severe: number analyzed (Participants) | 47 | 43 | 44 | 29 | 31 | 28
  Day 3: Severe | 17.0 | 18.6 | 9.1 | 6.9 | 12.9 | 10.7
  Day 3: Very severe: number analyzed (Participants) | 47 | 43 | 44 | 29 | 31 | 28
  Day 3: Very severe | 6.4 | 2.3 | 4.5 | 0 | 0 | 0
  Day 5: None: number analyzed (Participants) | 47 | 43 | 43 | 30 | 32 | 28
  Day 5: None | 2.1 | 0 | 7.0 | 3.3 | 0 | 3.6
  Day 5: Very mild: number analyzed (Participants) | 47 | 43 | 43 | 30 | 32 | 28
  Day 5: Very mild | 23.4 | 23.3 | 16.3 | 10.0 | 12.5 | 10.7
  Day 5: Mild: number analyzed (Participants) | 47 | 43 | 43 | 30 | 32 | 28
  Day 5: Mild | 38.3 | 27.9 | 32.6 | 36.7 | 43.8 | 32.1
  Day 5: Moderate: number analyzed (Participants) | 47 | 43 | 43 | 30 | 32 | 28
  Day 5: Moderate | 21.3 | 39.5 | 41.9 | 46.7 | 43.8 | 46.4
  Day 5: Severe: number analyzed (Participants) | 47 | 43 | 43 | 30 | 32 | 28
  Day 5: Severe | 10.6 | 9.3 | 2.3 | 3.3 | 0 | 7.1
  Day 5: Very severe: number analyzed (Participants) | 47 | 43 | 43 | 30 | 32 | 28
  Day 5: Very severe | 4.3 | 0 | 0 | 0 | 0 | 0
  Day 8: None: number analyzed (Participants) | 46 | 43 | 42 | 31 | 33 | 27
  Day 8: None | 13.0 | 16.3 | 26.2 | 12.9 | 6.1 | 7.4
  Day 8: Very mild: number analyzed (Participants) | 46 | 43 | 42 | 31 | 33 | 27
  Day 8: Very mild | 30.4 | 37.2 | 28.6 | 35.5 | 45.5 | 25.9
  Day 8: Mild: number analyzed (Participants) | 46 | 43 | 42 | 31 | 33 | 27
  Day 8: Mild | 34.8 | 23.3 | 28.6 | 38.7 | 27.3 | 48.1
  Day 8: Moderate: number analyzed (Participants) | 46 | 43 | 42 | 31 | 33 | 27
  Day 8: Moderate | 17.4 | 23.3 | 16.7 | 12.9 | 21.2 | 14.8
  Day 8: Severe: number analyzed (Participants) | 46 | 43 | 42 | 31 | 33 | 27
  Day 8: Severe | 2.2 | 0 | 0 | 0 | 0 | 0
  Day 8: Very severe: number analyzed (Participants) | 46 | 43 | 42 | 31 | 33 | 27
  Day 8: Very severe | 2.2 | 0 | 0 | 0 | 0 | 3.7
  Day 14: None: number analyzed (Participants) | 41 | 40 | 41 | 30 | 30 | 28
  Day 14: None | 48.8 | 55.0 | 58.5 | 70.0 | 63.3 | 67.9
  Day 14: Very mild: number analyzed (Participants) | 41 | 40 | 41 | 30 | 30 | 28
  Day 14: Very mild | 36.6 | 30.0 | 26.8 | 20.0 | 13.3 | 17.9
  Day 14: Mild: number analyzed (Participants) | 41 | 40 | 41 | 30 | 30 | 28
  Day 14: Mild | 12.2 | 2.5 | 7.3 | 6.7 | 16.7 | 10.7
  Day 14: Moderate: number analyzed (Participants) | 41 | 40 | 41 | 30 | 30 | 28
  Day 14: Moderate | 2.4 | 10.0 | 7.3 | 3.3 | 6.7 | 0
  Day 14: Severe: number analyzed (Participants) | 41 | 40 | 41 | 30 | 30 | 28
  Day 14: Severe | 0 | 2.5 | 0 | 0 | 0 | 3.6
  Day 14: Very severe: number analyzed (Participants) | 41 | 40 | 41 | 30 | 30 | 28
  Day 14: Very severe | 0 | 0 | 0 | 0 | 0 | 0
  Day 21: None: number analyzed (Participants) | 27 | 37 | 33 | 25 | 24 | 22
  Day 21: None | 66.7 | 67.6 | 57.6 | 84.0 | 83.3 | 86.4
  Day 21: Very mild: number analyzed (Participants) | 27 | 37 | 33 | 25 | 24 | 22
  Day 21: Very mild | 18.5 | 18.9 | 24.2 | 8.0 | 12.5 | 4.5
  Day 21: Mild: number analyzed (Participants) | 27 | 37 | 33 | 25 | 24 | 22
  Day 21: Mild | 11.1 | 2.7 | 12.1 | 0 | 4.2 | 9.1
  Day 21: Moderate: number analyzed (Participants) | 27 | 37 | 33 | 25 | 24 | 22
  Day 21: Moderate | 3.7 | 8.1 | 6.1 | 8.0 | 0 | 0
  Day 21: Severe: number analyzed (Participants) | 27 | 37 | 33 | 25 | 24 | 22
  Day 21: Severe | 0 | 2.7 | 0 | 0 | 0 | 0
  Day 21: Very severe: number analyzed (Participants) | 27 | 37 | 33 | 25 | 24 | 22
  Day 21: Very severe | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Percentage of Participants by Health Status Assessment Based on PRESORS Caregiver (ObsRO) General Question Over Time
Description: Percentage of participants by health status assessment based on PRESORS caregiver (ObsRO) general question over time was assessed. PRESORS is a questionnaire recording presence and severity of signs and symptoms of RSV disease (fever, cough, sputum, wheezing, difficulty breathing, nasal congestion, and feeding issues). Health status was assessed by a question (how is the child's health now) of PRESORS questionnaire and responses were categorized as: 1) excellent, 2) very good, 3) good, 4) fair, 5) poor, and 6) very poor.
Time Frame: Baseline, Days 3, 5, 8, 14, and 21
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44 | 32 | 33 | 28
Percentage of participants
  Baseline: Excellent: number analyzed (Participants) | 45 | 43 | 41 | 28 | 27 | 26
  Baseline: Excellent | 0 | 2.3 | 0 | 0 | 3.7 | 0
  Baseline: Very good: number analyzed (Participants) | 45 | 43 | 41 | 28 | 27 | 26
  Baseline: Very good | 0 | 4.7 | 0 | 3.6 | 0 | 7.7
  Baseline: Good: number analyzed (Participants) | 45 | 43 | 41 | 28 | 27 | 26
  Baseline: Good | 4.4 | 7.0 | 7.3 | 14.3 | 11.1 | 3.8
  Baseline: Fair: number analyzed (Participants) | 45 | 43 | 41 | 28 | 27 | 26
  Baseline: Fair | 42.2 | 51.2 | 43.9 | 57.1 | 40.7 | 23.1
  Baseline: Poor: number analyzed (Participants) | 45 | 43 | 41 | 28 | 27 | 26
  Baseline: Poor | 48.9 | 30.2 | 48.8 | 25.0 | 44.4 | 65.4
  Baseline: Very poor: number analyzed (Participants) | 45 | 43 | 41 | 28 | 27 | 26
  Baseline: Very poor | 4.4 | 4.7 | 0 | 0 | 0 | 0
  Day 3: Excellent: number analyzed (Participants) | 47 | 44 | 43 | 29 | 31 | 28
  Day 3: Excellent | 0 | 0 | 0 | 3.4 | 0 | 0
  Day 3: Very good: number analyzed (Participants) | 47 | 44 | 43 | 29 | 31 | 28
  Day 3: Very good | 8.5 | 9.3 | 2.3 | 0 | 0 | 0
  Day 3: Good: number analyzed (Participants) | 47 | 44 | 43 | 29 | 31 | 28
  Day 3: Good | 23.4 | 20.9 | 34.1 | 17.2 | 12.9 | 10.7
  Day 3: Fair: number analyzed (Participants) | 47 | 44 | 43 | 29 | 31 | 28
  Day 3: Fair | 38.3 | 46.5 | 45.5 | 58.6 | 41.9 | 53.6
  Day 3: Poor: number analyzed (Participants) | 47 | 44 | 43 | 29 | 31 | 28
  Day 3: Poor | 21.3 | 23.3 | 13.6 | 20.7 | 45.2 | 35.7
  Day 3: Very poor: number analyzed (Participants) | 47 | 44 | 43 | 29 | 31 | 28
  Day 3: Very poor | 8.5 | 0 | 4.5 | 0 | 0 | 0
  Day 5: Excellent: number analyzed (Participants) | 47 | 43 | 43 | 30 | 32 | 28
  Day 5: Excellent | 2.1 | 0 | 0 | 6.7 | 0 | 0
  Day 5: Very good: number analyzed (Participants) | 47 | 43 | 43 | 30 | 32 | 28
  Day 5: Very good | 19.1 | 9.3 | 20.9 | 0 | 6.3 | 3.6
  Day 5: Good: number analyzed (Participants) | 47 | 43 | 43 | 30 | 32 | 28
  Day 5: Good | 23.4 | 41.9 | 37.2 | 26.7 | 31.3 | 28.6
  Day 5: Fair: number analyzed (Participants) | 47 | 43 | 43 | 30 | 32 | 28
  Day 5: Fair | 36.2 | 39.5 | 34.9 | 63.3 | 40.6 | 42.9
  Day 5: Poor: number analyzed (Participants) | 47 | 43 | 43 | 30 | 32 | 28
  Day 5: Poor | 12.8 | 9.3 | 7.0 | 3.3 | 21.9 | 25.0
  Day 5: Very poor: number analyzed (Participants) | 47 | 43 | 43 | 30 | 32 | 28
  Day 5: Very poor | 6.4 | 0 | 0 | 0 | 0 | 0
  Day 8: Excellent: number analyzed (Participants) | 46 | 43 | 42 | 31 | 33 | 27
  Day 8: Excellent | 13.0 | 9.3 | 16.7 | 6.5 | 3.0 | 3.7
  Day 8: Very good: number analyzed (Participants) | 46 | 43 | 42 | 31 | 33 | 27
  Day 8: Very good | 23.9 | 32.6 | 21.4 | 19.4 | 21.2 | 22.2
  Day 8: Good: number analyzed (Participants) | 46 | 43 | 42 | 31 | 33 | 27
  Day 8: Good | 32.6 | 32.6 | 38.1 | 48.4 | 36.4 | 33.3
  Day 8: Fair: number analyzed (Participants) | 46 | 43 | 42 | 31 | 33 | 27
  Day 8: Fair | 23.9 | 25.6 | 21.4 | 22.6 | 36.4 | 33.3
  Day 8: Poor: number analyzed (Participants) | 46 | 43 | 42 | 31 | 33 | 27
  Day 8: Poor | 4.3 | 0 | 2.4 | 3.2 | 3.0 | 3.7
  Day 8: Very poor: number analyzed (Participants) | 46 | 43 | 42 | 31 | 33 | 27
  Day 8: Very poor | 2.2 | 0 | 0 | 0 | 0 | 3.7
  Day 14: Excellent: number analyzed (Participants) | 41 | 40 | 41 | 30 | 30 | 28
  Day 14: Excellent | 24.4 | 42.5 | 43.9 | 50.0 | 56.7 | 53.6
  Day 14: Very good: number analyzed (Participants) | 41 | 40 | 41 | 30 | 30 | 28
  Day 14: Very good | 43.9 | 47.5 | 36.6 | 23.3 | 16.7 | 28.6
  Day 14: Good: number analyzed (Participants) | 41 | 40 | 41 | 30 | 30 | 28
  Day 14: Good | 19.5 | 5.0 | 9.8 | 20.0 | 16.7 | 7.1
  Day 14: Fair: number analyzed (Participants) | 41 | 40 | 41 | 30 | 30 | 28
  Day 14: Fair | 9.8 | 5.0 | 7.3 | 6.7 | 6.7 | 3.6
  Day 14: Poor: number analyzed (Participants) | 41 | 40 | 41 | 30 | 30 | 28
  Day 14: Poor | 2.4 | 0 | 2.4 | 0 | 3.3 | 3.6
  Day 14: Very poor: number analyzed (Participants) | 41 | 40 | 41 | 30 | 30 | 28
  Day 14: Very poor | 0 | 0 | 0 | 0 | 0 | 3.6
  Day 21: Excellent: number analyzed (Participants) | 27 | 37 | 33 | 25 | 24 | 22
  Day 21: Excellent | 55.6 | 45.9 | 45.5 | 60.0 | 79.2 | 68.2
  Day 21: Very good: number analyzed (Participants) | 27 | 37 | 33 | 25 | 24 | 22
  Day 21: Very good | 22.2 | 32.4 | 33.3 | 28.0 | 12.5 | 9.1
  Day 21: Good: number analyzed (Participants) | 27 | 37 | 33 | 25 | 24 | 22
  Day 21: Good | 11.1 | 13.5 | 15.2 | 8.0 | 4.2 | 13.6
  Day 21: Fair: number analyzed (Participants) | 27 | 37 | 33 | 25 | 24 | 22
  Day 21: Fair | 11.1 | 5.4 | 6.1 | 0 | 4.2 | 9.1
  Day 21: Poor: number analyzed (Participants) | 27 | 37 | 33 | 25 | 24 | 22
  Day 21: Poor | 0 | 2.7 | 0 | 4.0 | 0 | 0
  Day 21: Very poor: number analyzed (Participants) | 27 | 37 | 33 | 25 | 24 | 22
  Day 21: Very poor | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Percentage of Participants With Worsening or Improvement Status of RSV Disease
Description: Percentage of participants with worsening or improvement of RSV disease based on general questions of overall health was assessed. Improvement or worsening was assessed by a question 'Would you say the child's RSV symptoms have improved, are about the same or are worse than when the child entered the study' and responses were categorized as: 1) very much improved, 2) much improved, 3) a little improved, 4) about the same, 5) a little worse, 6) much worse, and 7) very much worse".
Time Frame: Days 14 and 21
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44 | 32 | 33 | 28
Percentage of participants
  Day 14: Very much improved: number analyzed (Participants) | 41 | 40 | 40 | 30 | 29 | 28
  Day 14: Very much improved | 58.5 | 57.5 | 67.5 | 76.7 | 51.7 | 64.3
  Day 14: Much improved: number analyzed (Participants) | 41 | 40 | 40 | 30 | 29 | 28
  Day 14: Much improved | 34.1 | 40.0 | 30.0 | 20.0 | 37.9 | 32.1
  Day 14: A little improved: number analyzed (Participants) | 41 | 40 | 40 | 30 | 29 | 28
  Day 14: A little improved | 7.3 | 2.5 | 2.5 | 0 | 3.4 | 0
  Day 14: About the same: number analyzed (Participants) | 41 | 40 | 40 | 30 | 29 | 28
  Day 14: About the same | 0 | 0 | 0 | 3.3 | 3.4 | 3.6
  Day 14: A little worse: number analyzed (Participants) | 41 | 40 | 40 | 30 | 29 | 28
  Day 14: A little worse | 0 | 0 | 0 | 0 | 3.4 | 0
  Day 14: Much worse: number analyzed (Participants) | 41 | 40 | 40 | 30 | 29 | 28
  Day 14: Much worse | 0 | 0 | 0 | 0 | 0 | 0
  Day 14: Very much worse: number analyzed (Participants) | 41 | 40 | 40 | 30 | 29 | 28
  Day 14: Very much worse | 0 | 0 | 0 | 0 | 0 | 0
  Day 21: Very much improved: number analyzed (Participants) | 27 | 36 | 32 | 25 | 23 | 22
  Day 21: Very much improved | 77.8 | 63.9 | 56.3 | 76.0 | 78.3 | 77.3
  Day 21: Much improved: number analyzed (Participants) | 27 | 36 | 32 | 25 | 23 | 22
  Day 21: Much improved | 14.8 | 30.6 | 37.5 | 24.0 | 21.7 | 13.6
  Day 21: A little improved: number analyzed (Participants) | 27 | 36 | 32 | 25 | 23 | 22
  Day 21: A little improved | 3.7 | 2.8 | 3.1 | 0 | 0 | 0
  Day 21: About the same: number analyzed (Participants) | 27 | 36 | 32 | 25 | 23 | 22
  Day 21: About the same | 3.7 | 2.8 | 3.1 | 0 | 0 | 0
  Day 21: A little worse: number analyzed (Participants) | 27 | 36 | 32 | 25 | 23 | 22
  Day 21: A little worse | 0 | 0 | 0 | 0 | 0 | 9.1
  Day 21: Much worse: number analyzed (Participants) | 27 | 36 | 32 | 25 | 23 | 22
  Day 21: Much worse | 0 | 0 | 0 | 0 | 0 | 0
  Day 21: Very much worse: number analyzed (Participants) | 27 | 36 | 32 | 25 | 23 | 22
  Day 21: Very much worse | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Percentage of Participants by Return to Pre-RSV Disease Health Status Assessment Based on PRESORS Caregiver (ObsRO) General Question Over Time
Description: Percentage of participants by return to pre-RSV disease health status assessment based on PRESORS caregiver (ObsRO) general question over time was assessed by a question (Has the child's health returned to normal [how it was before RSV?]) of PRESORS questionnaire and responses were categorized as: 1) No, and 2) Yes. PRESORS is a questionnaire recording presence and severity of signs and symptoms of RSV disease (fever, cough, sputum, wheezing, difficulty breathing, nasal congestion, and feeding issues). Below results are reported for category 'Yes'.
Time Frame: Baseline, Days 3, 5, 8, 14, and 21
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44 | 32 | 33 | 28
Percentage of participants
  Baseline: number analyzed (Participants) | 11 | 4 | 9 | 9 | 9 | 8
  Baseline | 0 | 0 | 0 | 22.2 | 0 | 12.5
  Day 3: number analyzed (Participants) | 39 | 35 | 32 | 25 | 25 | 23
  Day 3 | 15.4 | 8.6 | 28.1 | 12.0 | 12.0 | 4.3
  Day 5: number analyzed (Participants) | 42 | 37 | 39 | 25 | 23 | 23
  Day 5 | 23.8 | 16.2 | 25.6 | 16.0 | 4.3 | 0
  Day 8: number analyzed (Participants) | 40 | 38 | 34 | 27 | 25 | 20
  Day 8 | 37.5 | 44.7 | 58.8 | 51.9 | 36.0 | 10.0
  Day 14: number analyzed (Participants) | 29 | 36 | 32 | 27 | 21 | 26
  Day 14 | 72.4 | 77.8 | 84.4 | 81.5 | 85.7 | 73.1
  Day 21: number analyzed (Participants) | 27 | 36 | 32 | 25 | 23 | 22
  Day 21 | 81.5 | 86.1 | 84.4 | 92.0 | 95.7 | 95.5

15. Secondary Outcome: Respiratory Rate (RR) Over Time
Description: Respiratory rate (RR) was measured by the investigator over time.
Time Frame: Baseline, Days 3, 5, 8, 14 and 21
Population: The Safety analysis set included all participants who received at least 1 dose of study agent, and were analyzed as treated, regardless of the randomized treatment group assigned. Here, 'n' (number analyzed) represents number of participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: Breaths/minute
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31
Breaths/minute
  Baseline | 45.0 (10.60) | 45.6 (11.82) | 45.7 (10.85) | 41.3 (13.66) | 41.3 (11.76) | 37.0 (8.77)
  Day 3: number analyzed (Participants) | 48 | 48 | 48 | 33 | 34 | 31
  Day 3 | 44.1 (11.44) | 41.8 (10.13) | 42.7 (10.04) | 37.9 (10.16) | 37.3 (9.54) | 34.4 (9.19)
  Day 5: number analyzed (Participants) | 47 | 45 | 46 | 33 | 34 | 31
  Day 5 | 38.3 (9.36) | 38.1 (9.57) | 39.1 (8.81) | 38.2 (13.37) | 38.1 (8.89) | 35.4 (9.53)
  Day 8: number analyzed (Participants) | 47 | 44 | 46 | 32 | 34 | 31
  Day 8 | 35.5 (7.90) | 34.4 (7.87) | 39.2 (9.45) | 37.4 (11.70) | 36.9 (9.75) | 34.0 (10.54)
  Day 14: number analyzed (Participants) | 47 | 45 | 46 | 30 | 32 | 29
  Day 14 | 35.6 (7.13) | 34.9 (8.89) | 35.2 (7.45) | 35.7 (9.27) | 35.6 (10.53) | 32.6 (8.38)
  Day 21: number analyzed (Participants) | 46 | 48 | 44 | 31 | 34 | 31
  Day 21 | 36.07 (10.21) | 34.9 (8.96) | 36.6 (7.43) | 36.4 (9.61) | 35.5 (9.65) | 34.7 (11.09)

16. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Change from baseline in respiratory rate was derived based on the reported measurements of respiratory rate over time. The respiratory rate over time was reported by the investigator.
Time Frame: Baseline to Days 3, 5, 8, 14 and 21
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Breaths/minute
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31
Breaths/minute
  Day 3: number analyzed (Participants) | 48 | 48 | 48 | 33 | 34 | 31
  Day 3 | -0.8 (10.88) | -3.5 (11.99) | -3.0 (12.43) | -3.7 (12.47) | -4.0 (9.54) | -2.6 (9.20)
  Day 5: number analyzed (Participants) | 47 | 45 | 46 | 33 | 34 | 31
  Day 5 | -6.5 (9.41) | -7.1 (11.13) | -7.0 (11.94) | -3.4 (8.59) | -3.3 (8.40) | -1.5 (9.62)
  Day 8: number analyzed (Participants) | 47 | 44 | 46 | 32 | 34 | 31
  Day 8 | -9.4 (9.19) | -11.4 (12.96) | -6.3 (12.69) | -4.4 (11.56) | -4.4 (10.39) | -2.9 (10.54)
  Day 14: number analyzed (Participants) | 47 | 45 | 46 | 30 | 32 | 29
  Day 14 | -9.3 (9.96) | -10.3 (12.59) | -10.2 (10.92) | -6.4 (3.13) | -5.8 (12.82) | -4.0 (9.92)
  Day 21: number analyzed (Participants) | 46 | 48 | 44 | 31 | 34 | 31
  Day 21 | -8.4 (10.84) | -10.4 (13.01) | -9.8 (12.36) | -5.5 (14.15) | -5.8 (11.95) | -2.3 (13.25)

17. Secondary Outcome: Heart Rate Over Time
Description: Heart rate was measured by the investigator over time.
Time Frame: Baseline, Days 3, 5, 8, 14 and 21
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31
Beats/minute
  Baseline | 143.2 (17.40) | 138.9 (17.57) | 139.0 (18.57) | 131.2 (24.28) | 135.6 (19.35) | 126.1 (22.55)
  Day 3: number analyzed (Participants) | 48 | 48 | 48 | 33 | 34 | 31
  Day 3 | 138.8 (16.82) | 137.5 (18.25) | 138.5 (17.06) | 127.8 (20.99) | 128.3 (17.97) | 118.8 (28.10)
  Day 5: number analyzed (Participants) | 47 | 46 | 47 | 33 | 34 | 31
  Day 5 | 136.0 (15.81) | 132.7 (18.28) | 16.1 (19.68) | 119.2 (14.75) | 122.6 (19.85) | 120.4 (23.31)
  Day 8: number analyzed (Participants) | 48 | 44 | 46 | 32 | 34 | 31
  Day 8 | 133.3 (17.59) | 127.9 (18.13) | 134.0 (19.14) | 118.7 (20.25) | 120.0 (19.61) | 118.9 (27.04)
  Day 14: number analyzed (Participants) | 47 | 45 | 46 | 30 | 32 | 29
  Day 14 | 131.7 (19.81) | 132.4 (19.33) | 134.4 (20.70) | 117.4 (18.17) | 118.0 (19.17) | 115.2 (18.82)
  Day 21: number analyzed (Participants) | 46 | 48 | 44 | 31 | 34 | 31
  Day 21 | 128.2 (20.27) | 131.5 (15.74) | 132.5 (19.14) | 117.2 (22.56) | 125.3 (20.95) | 115.2 (19.78)

18. Secondary Outcome: Change From Baseline in Heart Rate
Description: Change from baseline in heart rate was assessed.
Time Frame: Baseline to Days 3, 5, 8, 14 and 21
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31
Beats/minute
  Day 3: number analyzed (Participants) | 48 | 48 | 48 | 33 | 34 | 31
  Day 3 | -4.9 (19.36) | -1.6 (19.82) | -0.6 (18.84) | -3.0 (24.71) | -7.4 (16.83) | -7.3 (28.39)
  Day 5: number analyzed (Participants) | 47 | 46 | 47 | 33 | 34 | 31
  Day 5 | -7.9 (20.31) | -5.8 (22.94) | -2.9 (20.56) | -11.6 (18.55) | -13.0 (17.11) | -5.6 (28.53)
  Day 8: number analyzed (Participants) | 48 | 44 | 46 | 32 | 34 | 31
  Day 8 | -10.4 (18.45) | -12.2 (23.20) | -5.2 (22.02) | -12.7 (26.09) | -15.6 (20.67) | -7.2 (35.90)
  Day 14: number analyzed (Participants) | 47 | 45 | 46 | 30 | 32 | 29
  Day 14 | -12.0 (21.79) | -6.5 (23.99) | -5.1 (22.44) | -14.4 (24.62) | -17.7 (17.69) | -10.1 (28.02)
  Day 21: number analyzed (Participants) | 46 | 48 | 44 | 31 | 34 | 31
  Day 21 | -15.0 (23.80) | -7.7 (25.88) | -6.5 (19.52) | -14.0 (25.38) | -10.4 (21.02) | -10.9 (28.63)

19. Secondary Outcome: Body Temperature Over Time
Description: Body temperature was reported over time (either investigator or caregiver measured).
Time Frame: Baseline, Days 3, 5, 8, 14 and 21
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Degrees celsius
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31
Degrees celsius
  Baseline | 36.84 (0.635) | 36.64 (0.468) | 36.82 (0.623) | 36.84 (0.613) | 36.94 (0.845) | 36.79 (0.785)
  Day 3: number analyzed (Participants) | 48 | 48 | 48 | 33 | 34 | 31
  Day 3 | 36.77 (0.464) | 36.87 (0.524) | 36.80 (0.601) | 37.14 (0.725) | 37.20 (0.694) | 36.98 (0.817)
  Day 5: number analyzed (Participants) | 49 | 48 | 48 | 33 | 34 | 31
  Day 5 | 36.75 (0.407) | 36.54 (0.557) | 36.70 (0.408) | 36.87 (0.567) | 36.71 (0.348) | 36.84 (0.718)
  Day 8: number analyzed (Participants) | 48 | 47 | 48 | 33 | 34 | 31
  Day 8 | 36.70 (0.416) | 36.73 (0.513) | 36.65 (0.441) | 36.67 (0.369) | 36.76 (0.536) | 36.74 (0.559)
  Day 14: number analyzed (Participants) | 47 | 45 | 47 | 33 | 34 | 31
  Day 14 | 36.86 (0.315) | 36.68 (0.440) | 36.60 (0.396) | 36.63 (0.357) | 36.72 (0.364) | 36.59 (0.377)
  Day 21: number analyzed (Participants) | 47 | 48 | 47 | 33 | 34 | 31
  Day 21 | 36.76 (0.577) | 36.67 (0.407) | 36.66 (0.573) | 36.74 (0.615) | 36.64 (0.292) | 36.62 (0.418)

20. Secondary Outcome: Change From Baseline in Body Temperature
Description: Change from baseline in body temperature (either investigator or caregiver measured) was assessed.
Time Frame: Baseline to Days 3, 5, 8, 14 and 21
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Degrees celsius
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31
Degrees celsius
  Day 3: number analyzed (Participants) | 48 | 48 | 48 | 33 | 34 | 30
  Day 3 | -0.08 (0.697) | 0.23 (0.541) | -0.02 (0.629) | 0.33 (0.768) | 0.26 (0.835) | 0.21 (0.724)
  Day 5: number analyzed (Participants) | 49 | 48 | 48 | 33 | 34 | 30
  Day 5 | -0.10 (0.713) | -0.09 (0.532) | -0.12 (0.627) | 0.07 (0.700) | -0.22 (0.767) | -0.04 (0.627)
  Day 8: number analyzed (Participants) | 48 | 47 | 48 | 33 | 34 | 30
  Day 8 | -0.13 (0.659) | 0.10 (0.600) | -0.17 (0.596) | -0.13 (0.588) | -0.17 (1.016) | -0.11 (0.772)
  Day 14: number analyzed (Participants) | 47 | 45 | 47 | 33 | 34 | 30
  Day 14 | 0.01 (0.594) | 0.04 (0.528) | -0.21 (0.609) | -0.17 (0.687) | -0.21 (0.866) | -0.19 (0.843)
  Day 21: number analyzed (Participants) | 47 | 48 | 47 | 33 | 34 | 30
  Day 21 | -0.09 (0.758) | 0.03 (0.519) | -0.17 (0.724) | -0.06 (0.704) | -0.30 (0.826) | -0.18 (0.913)

21. Secondary Outcome: Peripheral Capillary Oxygen Saturation (SpO2) Over Time
Description: Peripheral capillary oxygen saturation was measured by the investigator over time.
Time Frame: Baseline, Days 3, 5, 8, 14 and 21
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percentage of SpO2
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31
Percentage of SpO2
  Baseline: number analyzed (Participants) | 50 | 49 | 48 | 32 | 32 | 30
  Baseline | 97.3 (2.47) | 96.5 (3.44) | 96.6 (2.10) | 96.8 (2.07) | 96.7 (1.91) | 95.9 (2.92)
  Day 3: number analyzed (Participants) | 47 | 48 | 48 | 31 | 32 | 29
  Day 3 | 96.8 (2.46) | 96.3 (2.72) | 96.0 (2.43) | 96.9 (1.77) | 96.3 (3.12) | 96.5 (2.96)
  Day 5: number analyzed (Participants) | 47 | 46 | 47 | 32 | 32 | 30
  Day 5 | 97.3 (1.67) | 96.8 (3.74) | 96.7 (2.25) | 96.9 (1.68) | 97.1 (2.12) | 97.1 (2.43)
  Day 8: number analyzed (Participants) | 46 | 44 | 46 | 30 | 32 | 30
  Day 8 | 97.3 (1.99) | 97.3 (2.47) | 97.5 (1.74) | 97.8 (1.48) | 97.4 (2.69) | 97.9 (1.83)
  Day 14: number analyzed (Participants) | 44 | 43 | 45 | 29 | 29 | 28
  Day 14 | 98.1 (1.42) | 98.3 (1.84) | 98.1 (1.64) | 98.6 (2.03) | 98.6 (1.53) | 98.4 (1.73)
  Day 21: number analyzed (Participants) | 45 | 47 | 43 | 30 | 32 | 30
  Day 21 | 98.4 (1.47) | 98.2 (1.80) | 98.0 (2.12) | 98.5 (1.74) | 98.7 (1.36) | 98.9 (1.25)

22. Secondary Outcome: Change From Baseline in Peripheral Capillary Oxygen Saturation (SpO2)
Description: Change from baseline in peripheral capillary oxygen saturation levels was derived based on reported values over time.
Time Frame: Baseline to Days 3, 5, 8, 14, and 21
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percentage of SpO2
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31
Percentage of SpO2
  Day 3: number analyzed (Participants) | 47 | 48 | 48 | 31 | 32 | 29
  Day 3 | -0.5 (2.93) | -0.2 (3.09) | -0.6 (2.72) | 0.2 (2.31) | -0.4 (2.45) | 0.7 (1.63)
  Day 5: number analyzed (Participants) | 47 | 46 | 47 | 31 | 32 | 30
  Day 5 | 0.0 (2.92) | 0.4 (2.93) | 0.1 (2.38) | 0.1 (2.49) | 0.4 (2.41) | 1.2 (2.54)
  Day 8: number analyzed (Participants) | 46 | 44 | 46 | 30 | 32 | 30
  Day 8 | 0.1 (3.02) | 0.9 (3.53) | 0.8 (2.47) | 0.9 (2.59) | 0.8 (2.86) | 2.0 (3.36)
  Day 14: number analyzed (Participants) | 44 | 43 | 45 | 29 | 29 | 28
  Day 14 | 1.0 (2.28) | 1.7 (3.08) | 1.4 (2.32) | 2.0 (2.72) | 1.8 (2.05) | 2.6 (3.06)
  Day 21: number analyzed (Participants) | 45 | 47 | 43 | 29 | 32 | 30
  Day 21 | 1.1 (2.45) | 1.7 (3.38) | 1.3 (2.40) | 1.8 (2.57) | 2.0 (2.12) | 3.0 (2.80)

23. Secondary Outcome: Percentage of Participants Who Required (re)Hospitalization During Treatment and Follow-up
Description: Percentage of participants who required (re)hospitalization during treatment and follow-up was assessed. Percentage of participants requiring re-hospitalization following the initial hospital discharge was assessed in Cohort 1 participants (hospitalized cohort) whilst percentage of participants requiring hospitalization after first dose of study drug was assessed in Cohort 2 participants (outpatient cohort).
Time Frame: Up to Day 28
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44 | 32 | 33 | 28
Percentage of participants | 6.4 | 4.3 | 2.3 | 6.3 | 6.1 | 14.3

24. Secondary Outcome: Cohort 1: Time to Return to Age-adjusted Normal Values for Vital Signs
Description: Time to return to age-adjusted normal values from first dose of study drug based on the reported vital signs (respiratory rate, heart rate, SpO2 >=92%, and SpO2 >=95%) values was assessed. As per the study protocol and study design, this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure is only reported for Cohort 1.
Time Frame: Up to Day 28
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44
Hours
  Respiratory Rate | 13.6 [0.001 to 70.10] | 20.0 [0.001 to 43.50] | 30.2 [0.001 to 84.50]
  Heart Rate | 37.3 [0.001 to 51.50] | 17.0 [0.001 to 67.50] | 10.2 [0.001 to 160.50]
  SpO2 >=92% on Room Air | 65.4 [30.30 to 95.10] | 86.6 [45.30 to 119.20] | 68.9 [42.40 to 105.50]
  SpO2 >=95% on Room Air | 71.3 [47.70 to 99.30] | 87.0 [47.80 to 120.00] | 92.5 [48.50 to 141.10]

25. Secondary Outcome: Cohort 1: Time to Discharge From Hospital
Description: Time to discharge from hospital was derived from the reported discharge date/time and from first dose date/time. As per the study protocol and study design, this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure is only reported for Cohort 1.
Time Frame: Up to Day 28
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44
Hours | 96.2 [88.80 to 118.00] | 95.3 [67.20 to 140.30] | 96.2 [72.10 to 144.90]

26. Secondary Outcome: Cohort 1: Percentage of Participants Who Required Admission to the Intensive Care Unit (ICU)
Description: Percentage of participants who required admission to the ICU was assessed. This outcome measure was applicable for those participants that were not in ICU before first dose of study drug. As per the study protocol and study design, this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure is only reported for Cohort 1.
Time Frame: Up to Day 21
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 42 | 44 | 39
Percentage of participants | 2.4 | 4.5 | 2.6

27. Secondary Outcome: Cohort 1: Duration of ICU Stay
Description: Duration of ICU stay was derived based on the reported admission/discharge date/time for ICU. Duration defined as total number of hours a participant was in ICU from first dose of study drug until study termination. As per the study protocol and study design, this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure is only reported for Cohort 1.
Time Frame: Up to Day 21
Population: ITT-i analysis set included all randomized participants who were admitted to ICU and received at least one dose of study drug and who had centrally confirmed RSV RNA viral load of >=1 log10 copies/mL above the LLOQ of the RSV RT-qPCR assay at baseline. Analyses on ITT-i set were performed as randomized. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 6 | 5 | 6
Hours | 238.22 (70.570) | 206.94 (204.940) | 127.72 (89.389)

28. Secondary Outcome: Cohort 1: Time to Clinical Stability Evaluated by the Investigator
Description: Time to clinical stability was derived based on vital signs(SpO2 >= 92%, SpO2 >=95% on room air) assessments and supplementation end dates as collected. Time to clinical stability=time from initiation of study treatment until time at which following criteria were met: Time to return to age-adjusted normal value for otherwise healthy, pre-RSV infection status for participant with risk factor for severe RSV disease,no more oxygen supplementation in otherwise healthy participant, participant with risk factor for severe RSV disease and no more IV administered/nasogastric tube feeding/hydration supplementation in otherwise healthy participant or pre-RSV status of IV/nasogastric tube feeding/hydration in participant with risk factor for severe RSV disease. As per protocol and study design,this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure is only reported for Cohort 1.
Time Frame: Up to Day 21
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44
Hours
  SpO2 >=92% on Room Air | 95.8 [63.50 to 165.80] | 123.3 [82.00 to 169.10] | 176.5 [77.80 to 309.50]
  SpO2 >=95% on Room Air | 95.8 [71.20 to 165.90] | 134.8 [82.00 to 311.50] | 180.5 [85.70 to 315.40]

29. Secondary Outcome: Cohort 1: Percentage of Participants Who Required Supplemental Oxygen
Description: Percentage of participants who required supplemental oxygen after first dose of study drug was reported. This parameter was only for participants that did not require oxygen supplementation before first dose of study drug. As per the study protocol and study design, this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure is only reported for Cohort 1.
Time Frame: Up to Day 21
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 14 | 12 | 7
Percentage of participants | 21.4 | 25.0 | 28.6

30. Secondary Outcome: Cohort 1: Duration of Supplemental Oxygen
Description: Duration of supplemental oxygen was assessed. Duration was defined as total number of hours a participant used supplemental oxygen from first dose of study drug until study termination. As per the study protocol and study design, this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure is only reported for Cohort 1.
Time Frame: Up to Day 28
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 34 | 38 | 38
Hours | 74.25 [1.0 to 337.3] | 74.60 [0.2 to 573.5] | 68.05 [1.2 to 348.5]

31. Secondary Outcome: Cohort 1: Percentage of Participants Who Required Non-invasive Mechanical Ventilation Support
Description: Percentage of participants who required non-invasive mechanical ventilation support (example: continuous positive airway pressure) after first dose of study drug was assessed. This parameter was only for participants who did not require non-invasive mechanical ventilation support before first dose of study drug. As per the study protocol and study design, this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure is only reported for Cohort 1.
Time Frame: Up to Day 21
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 45 | 44 | 38
Percentage of participants | 2.2 | 6.8 | 2.6

32. Secondary Outcome: Cohort 1: Percentage of Participants Who Required Invasive Mechanical Ventilation Support
Description: Percentage of participants who required invasive mechanical ventilation support (example: endotracheal-mechanical ventilation) after first dose of study drug was assessed. This parameter was only for participants who did not require invasive mechanical ventilation support before first dose of study drug. As per the study protocol and study design, this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure is only reported for Cohort 1.
Time Frame: Up to Day 21
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44
Percentage of participants | 4.3 | 2.1 | 2.3

33. Secondary Outcome: Cohort 1: Percentage of Participants Who Required Non-invasive Non-mechanical Ventilation Support
Description: Percentage of participants who required non-invasive non-mechanical ventilation support (example: nasal cannula) after first dose of study drug was assessed. This parameter was only for participants who did not require non-invasive non-mechanical ventilation support before first dose of study drug. As per the study protocol and study design, this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure is only reported for Cohort 1.
Time Frame: Up to Day 21
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 16 | 14 | 11
Percentage of participants | 31.3 | 35.7 | 45.5

34. Secondary Outcome: Cohort 1: Duration of Non-invasive Ventilation Support
Description: For the subset of participants who received non-invasive ventilation post dose, duration for non-invasive ventilation could not be derived by individual type as start/end dates and times were not collected in full to allow breakdown of duration derivation by ventilation type and only overall duration of oxygen supplementation (overall ventilation support) could be derived which is reported in the outcome measure "Duration of Supplemental Oxygen". As per the study protocol and study design, this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure could only have been reported for Cohort 1.
Time Frame: Up to Day 21
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had centrally confirmed RSV RNA viral load of >=1 log10 copies/mL above LLOQ of RSV RT-qPCR assay at baseline. Analyses on ITT-i set were performed as randomized. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represents number of participants who were evaluable at specified categories.
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 0 | 0 | 0

35. Secondary Outcome: Cohort 1: Duration of Invasive Ventilation Support
Description: For the subset of participants who received invasive ventilation post dose, duration for invasive ventilation could not be derived by individual type as start/end dates and times were not collected in full to allow breakdown of duration derivation by ventilation type and only overall duration of oxygen supplementation (overall ventilation support) could be derived which is reported in the outcome measure "Duration of Supplemental Oxygen". As per the study protocol and study design, this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure could only have been reported for Cohort 1.
Time Frame: Up to Day 21
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had centrally confirmed RSV RNA viral load of >=1 log10 copies/mL above LLOQ of RSV RT-qPCR assay at baseline. Analyses on ITT-i set were performed as randomized.
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 0 | 0 | 0

36. Secondary Outcome: Cohort 1: Time to End of Supplemental Oxygen up to 72 Hours From First Hospital Discharge
Description: Time to end of supplemental oxygen up to 72 hours from first hospital discharge was assessed. Time to end of supplemental oxygen was defined as time (hours) from first dose of study drug to last end date/time of any oxygen supplementation received, but within 72 hours following first hospital discharge. As per the study protocol and study design, this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure is only reported for Cohort 1.
Time Frame: Up to end of supplemental oxygen including supplemental oxygen within 72 hours after first hospital discharge (up to Day 28)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44
Hours | 58.1 [22.90 to 75.90] | 57.9 [35.30 to 85.50] | 63.0 [31.80 to 92.00]

37. Secondary Outcome: Cohort 1: Percentage of Participants Who Needed Hydration and/or Feeding by Intravenous (IV) Administration or Nasogastric Tube
Description: Percentage of participants who needed hydration and/or feeding by IV Administration or nasogastric tube after the first dose of study drug was assessed. This parameter was only for participants who didn't require supplemental feeding/hydration before first dose of study drug. As per the study protocol and study design, this outcome measure was planned to be analyzed for participants who were hospitalized only. Only participants in Cohort 1 were hospitalized, hence this outcome measure is only reported for Cohort 1.
Time Frame: Up to Day 28
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 32 | 32 | 26
Percentage of participants | 6.3 | 15.6 | 19.2

38. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Percentage of participants with adverse events was assessed. An AE is any untoward medical occurrence in clinical study participants administered a medicinal (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the intervention.
Time Frame: Up to Day 28
Population: The safety analysis set included all participants who received at least 1 dose of study agent, and were analyzed as treated, regardless of the randomized treatment group assigned.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31
Percentage of Participants | 58.0 | 59.2 | 64.6 | 47.1 | 58.8 | 41.9

39. Secondary Outcome: Percentage of Participants With Abnormal Laboratory Findings
Description: Percentage of participants with abnormal laboratory findings (chemistry and hematology) worst toxicity grade was assessed based on Division of Microbiology and Infectious Diseases (DMID) toxicity grading scale. DMID toxicity grades range from 1 to 4. Grade 1 = mild: transient or mild discomfort (<48 hours); no medical intervention/therapy required. Grade 2 = moderate: mild to moderate limitation in activity - some assistance may be needed; no or minimal medical intervention/therapy required. Grade 3 = severe: marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalizations possible. Grade 4 = life-threatening or death: Extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable.
Time Frame: Up to Day 28
Population: The Safety analysis set included all participants who received at least 1 dose of study agent, and were analyzed as treated, regardless of the randomized treatment group assigned. Here, 'n' (number analyzed) represents number of participants who were evaluable for the specified categories.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31
Percentage of Participants
  Chemistry: Alanine Transaminase (ALT): Grade 1: number analyzed (Participants) | 22 | 27 | 22 | 32 | 28 | 29
  Chemistry: Alanine Transaminase (ALT): Grade 1 | 13.6 | 0 | 0 | 0 | 3.6 | 3.4
  Chemistry: ALT: Grade 2: number analyzed (Participants) | 22 | 27 | 22 | 32 | 28 | 29
  Chemistry: ALT: Grade 2 | 0 | 0 | 4.5 | 0 | 0 | 0
  Chemistry: ALT: Grade 3: number analyzed (Participants) | 22 | 27 | 22 | 32 | 28 | 29
  Chemistry: ALT: Grade 3 | 4.5 | 0 | 0 | 0 | 0 | 0
  Chemistry: Aspartate Aminotransferase (AST): Grade 1: number analyzed (Participants) | 22 | 25 | 22 | 31 | 29 | 30
  Chemistry: Aspartate Aminotransferase (AST): Grade 1 | 0 | 0 | 4.5 | 0 | 0 | 3.3
  Chemistry: AST: Grade 3: number analyzed (Participants) | 22 | 25 | 22 | 31 | 29 | 30
  Chemistry: AST: Grade 3 | 4.5 | 0 | 0 | 0 | 0 | 0
  Chemistry: Hyperbilirubinemia: Grade 2: number analyzed (Participants) | 37 | 37 | 34 | 34 | 34 | 31
  Chemistry: Hyperbilirubinemia: Grade 2 | 2.7 | 0 | 0 | 0 | 0 | 0
  Chemistry: Hyperglycemia: Grade 1: number analyzed (Participants) | 22 | 26 | 23 | 32 | 29 | 30
  Chemistry: Hyperglycemia: Grade 1 | 13.6 | 0 | 4.3 | 6.3 | 3.4 | 10.0
  Chemistry: Hyperkalemia: Grade 1: number analyzed (Participants) | 22 | 27 | 23 | 32 | 29 | 30
  Chemistry: Hyperkalemia: Grade 1 | 59.1 | 22.2 | 39.1 | 21.9 | 55.2 | 36.7
  Chemistry: Hyperkalemia: Grade 2: number analyzed (Participants) | 22 | 27 | 23 | 32 | 29 | 30
  Chemistry: Hyperkalemia: Grade 2 | 0 | 0 | 4.3 | 3.1 | 3.4 | 3.3
  Chemistry: Hyperkalemia: Grade 4: number analyzed (Participants) | 22 | 27 | 23 | 32 | 29 | 30
  Chemistry: Hyperkalemia: Grade 4 | 0 | 0 | 8.7 | 0 | 0 | 0
  Chemistry: Hypernatremia: Grade 2: number analyzed (Participants) | 22 | 27 | 23 | 32 | 29 | 30
  Chemistry: Hypernatremia: Grade 2 | 4.5 | 3.7 | 0 | 3.1 | 3.4 | 3.3
  Chemistry: Hypernatremia: Grade 3: number analyzed (Participants) | 22 | 27 | 23 | 32 | 29 | 30
  Chemistry: Hypernatremia: Grade 3 | 4.5 | 0 | 0 | 0 | 0 | 0
  Chemistry: Hyperuricemia: Grade 1: number analyzed (Participants) | 22 | 27 | 23 | 34 | 34 | 31
  Chemistry: Hyperuricemia: Grade 1 | 0 | 0 | 4.3 | 0 | 0 | 0
  Chemistry: Hypoglycemia: Grade 1: number analyzed (Participants) | 22 | 26 | 23 | 32 | 29 | 30
  Chemistry: Hypoglycemia: Grade 1 | 4.5 | 0 | 4.3 | 6.3 | 3.4 | 0
  Chemistry: Hypomagnesemia: Grade 1: number analyzed (Participants) | 22 | 27 | 23 | 32 | 29 | 30
  Chemistry: Hypomagnesemia: Grade 1 | 0 | 3.7 | 4.3 | 3.1 | 0 | 0
  Chemistry: Hypomagnesemia: Grade 2: number analyzed (Participants) | 22 | 27 | 23 | 32 | 29 | 30
  Chemistry: Hypomagnesemia: Grade 2 | 0 | 0 | 4.3 | 0 | 0 | 0
  Chemistry: Hypomagnesemia: Grade 3: number analyzed (Participants) | 22 | 27 | 23 | 32 | 29 | 30
  Chemistry: Hypomagnesemia: Grade 3 | 0 | 0 | 4.3 | 0 | 0 | 0
  Chemistry: Hyponatremia: Grade 2: number analyzed (Participants) | 22 | 27 | 23 | 32 | 29 | 30
  Chemistry: Hyponatremia: Grade 2 | 4.5 | 3.7 | 0 | 0 | 0 | 10.0
  Hematology: Absolute Neutrophil Count: Grade 1: number analyzed (Participants) | 37 | 35 | 36 | 33 | 33 | 28
  Hematology: Absolute Neutrophil Count: Grade 1 | 13.5 | 11.4 | 2.8 | 3.0 | 9.1 | 0
  Hematology: Absolute Neutrophil Count: Grade 3: number analyzed (Participants) | 37 | 35 | 36 | 33 | 33 | 28
  Hematology: Absolute Neutrophil Count: Grade 3 | 0 | 2.9 | 0 | 0 | 0 | 0
  Hematology: Activated Partial Thromboplastin Time: Grade 1: number analyzed (Participants) | 9 | 10 | 15 | 1 | 3 | 3
  Hematology: Activated Partial Thromboplastin Time: Grade 1 | 11.1 | 0 | 0 | 0 | 0 | 33.3
  Hematology: Hemoglobin: Grade 1: number analyzed (Participants) | 38 | 36 | 35 | 34 | 34 | 31
  Hematology: Hemoglobin: Grade 1 | 7.9 | 5.6 | 2.9 | 0 | 0 | 0
  Hematology: Hemoglobin: Grade 2: number analyzed (Participants) | 38 | 36 | 35 | 34 | 34 | 31
  Hematology: Hemoglobin: Grade 2 | 2.6 | 2.8 | 0 | 0 | 0 | 0
  Hematology: Prothrombin Time: Grade 1: number analyzed (Participants) | 9 | 10 | 15 | 34 | 34 | 31
  Hematology: Prothrombin Time: Grade 1 | 0 | 10.0 | 0 | 0 | 0 | 0
  Hematology: Prothrombin Time: Grade 3: number analyzed (Participants) | 9 | 10 | 15 | 34 | 34 | 31
  Hematology: Prothrombin Time: Grade 3 | 11.1 | 0 | 6.7 | 0 | 0 | 0
  Chemistry: Hyperglycemia: Grade 2: number analyzed (Participants) | 22 | 26 | 23 | 32 | 29 | 30
  Chemistry: Hyperglycemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 3.3

40. Secondary Outcome: Percentage of Participants With Abnormal Electrocardiograms (ECGs) Findings
Description: Percentage of participants with abnormal ECG (PR interval [for age 0 to 2 years: >150 msec is abnormally high, for age group 2 to <3.5 years: <100 msec is abnormally low and >150 msec is abnormally high]; QRS interval [for 0 to 2 years: >79 msec is abnormally high, for age group 2 to <3.5 years: <40 msec is abnormally low and >79 msec is abnormally high]; QT interval [for age 0 to 2 years: >500 msec is abnormally high, for age group 2 to <18 years: <320 msec is abnormally low and >450 msec is abnormally high]; RR interval [for age 0 to 3 months: <333 msec is abnormally low and >750 msec is abnormally high; for age group 3 to 12 months: <400 msec is abnormally low and >860 msec is abnormally high; for age 1 to 2 years: <430 msec is abnormally low and >1000 msec is abnormally high; for age group 2 to <18 years: <600 msec is abnormally low and >1200 msec is abnormally high]) findings were assessed.
Time Frame: Up to Day 28
Population: The Safety analysis set included all participants who received at least 1 dose of study agent, and were analyzed as treated, regardless of the randomized treatment group assigned. Here, 'n' (number analyzed) represents number of participants who were evaluable for specified categories (per ECG parameters).
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31
Percentage of Participants
  QRS Duration: Abnormally High: number analyzed (Participants) | 49 | 48 | 48 | 33 | 33 | 31
  QRS Duration: Abnormally High | 4.1 | 4.2 | 4.2 | 6.1 | 6.1 | 9.7
  RR Interval: Abnormally Low: number analyzed (Participants) | 49 | 48 | 48 | 33 | 33 | 31
  RR Interval: Abnormally Low | 12.2 | 8.3 | 12.5 | 21.2 | 15.2 | 9.7
  PR Interval: Abnormally Low: number analyzed (Participants) | 49 | 48 | 48 | 33 | 33 | 31
  PR Interval: Abnormally Low | 0 | 2.1 | 2.1 | 0 | 3.0 | 0
  QT Interval: Abnormally Low: number analyzed (Participants) | 49 | 48 | 48 | 33 | 33 | 31
  QT Interval: Abnormally Low | 2.0 | 4.2 | 2.1 | 3.0 | 9.1 | 3.2

41. Secondary Outcome: Percentage of Participants With Categorized Change From Baseline in ECG Parameters (QT, QTcB, QTcF)
Description: Percentage of participants with categorized change from Baseline in ECG parameters (QT/ QTcB/ QTcF interval) was assessed. Abnormal ECG change from baseline in QTc and QTcB Interval is categorized as borderline QTc change: 30 ms (milliseconds) to <60 ms, and abnormally high QTc change: greater than [>] 60 ms), and QTcF Interval is categorized as borderline QTc change: 30 ms to <60 ms, and abnormally high QTc change: >60 ms.
Time Frame: Baseline to Day 28
Population: The Safety analysis set included all participants who received at least 1 dose of study agent, and were analyzed as treated, regardless of the randomized treatment group assigned. Here, 'n' (number analyzed) represents number of participants who were evaluable per ECG parameter.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31
Percentage of participants
  QT Interval: Normal QT change: number analyzed (Participants) | 48 | 48 | 48 | 33 | 33 | 29
  QT Interval: Normal QT change | 66.7 | 70.8 | 68.8 | 66.7 | 57.6 | 58.6
  QT Interval: Borderline QT change: number analyzed (Participants) | 48 | 48 | 48 | 33 | 33 | 29
  QT Interval: Borderline QT change | 29.2 | 25.0 | 27.1 | 27.3 | 33.3 | 37.9
  QT Interval: Abnormally high QT change: number analyzed (Participants) | 48 | 48 | 48 | 33 | 33 | 29
  QT Interval: Abnormally high QT change | 4.2 | 4.2 | 4.2 | 6.1 | 9.1 | 3.4
  QTcB Interval: Normal QTc change: number analyzed (Participants) | 48 | 48 | 48 | 33 | 33 | 29
  QTcB Interval: Normal QTc change | 83.8 | 87.5 | 93.8 | 90.9 | 90.9 | 93.1
  QTcB Interval: Borderline QTc change: number analyzed (Participants) | 48 | 48 | 48 | 33 | 33 | 29
  QTcB Interval: Borderline QTc change | 14.6 | 12.5 | 6.3 | 9.1 | 9.1 | 6.9
  QTcB Interval: Abnormally high QTc change: number analyzed (Participants) | 48 | 48 | 48 | 33 | 33 | 29
  QTcB Interval: Abnormally high QTc change | 2.1 | 0 | 0 | 0 | 0 | 0
  QTcF Interval: Normal QTc change: number analyzed (Participants) | 48 | 48 | 48 | 33 | 33 | 29
  QTcF Interval: Normal QTc change | 81.3 | 83.3 | 83.3 | 90.9 | 78.8 | 86.3
  QTcF Interval: Borderline QTc change: number analyzed (Participants) | 48 | 48 | 48 | 33 | 33 | 29
  QTcF Interval: Borderline QTc change | 16.7 | 16.7 | 16.7 | 9.1 | 21.2 | 13.8
  QTcF Interval: Abnormally high QTc change: number analyzed (Participants) | 48 | 48 | 48 | 33 | 33 | 29
  QTcF Interval: Abnormally high QTc change | 2.1 | 0 | 0 | 0 | 0 | 0

42. Secondary Outcome: Percentage of Participants With Vital Signs Abnormalities
Description: Percentage of participants with vital signs (SBP,DBP, pulse rate, respiratory rate, body temperature and SpO2) abnormalities (abnormally low [ABL] and abnormally high [ABH]) were reported. DBP: ABL: <35 mmHg:0-3 months (mths), <40 mmHg:3 mths- <3.5 years,ABH: >65 mmHg:0-3 mths, >85 mmHg:3-12 mths, >90 mmHg:1-2 years, >70 mmHg: 2- <3.5 years; SBP:ABL: <60 mmHg:0-12 mths,<75 mmHg:1-2 years, <80:2- <3.5 years,ABH: >110:0-12 mths, >120 mmHg:1-2 years, >10 mmHg:2- <3.5 years; Pulse rate:ABL: <80 bpm:0-3 mths, <70 bpm:3 mths-12 mth,<60 bpm:1-2 years, <90 bpm:2- <3.5 years,ABH: >180 bpm:0-3 mths, >150 bpm:3 mths-12 mths, >140 bpm:1-2 years, >130:2- <3.5 years; Respiratory rate:ABL: <25 bpm:0-3 mths, <20 bpm: 3 mths-12 mths,<18 bpm:1-2 years, <20 bpm:2- <3.5 years, ABH:>70 bpm:0-3 mths, >60 bpm:3 mths-12 mths, >50 bpm:1-2 years, >35 bpm:2- <3.5 years; SpO2: ABL: <92%: 0-<3.5 years; Temperature (Celsius): ABH:>37.8:Tympanic, >38.0:forehead, oral, axillary, >37.2:rectal.
Time Frame: Up to Day 28
Population: The Safety analysis set included all participants who received at least 1 dose of study agent, and were analyzed as treated, regardless of the randomized treatment group assigned. Here, 'n' (number analyzed) represents number of participants evaluable per vital sign parameter. As per change in planned analysis, the upper limit for the last age group was 3.5 years instead of 3 years.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 50 | 49 | 48 | 34 | 34 | 31
Percentage of Participants
  Systolic Blood Pressure (SBP): Abnormally Low: number analyzed (Participants) | 49 | 48 | 48 | 33 | 34 | 31
  Systolic Blood Pressure (SBP): Abnormally Low | 2.0 | 2.1 | 8.3 | 12.1 | 8.8 | 9.7
  SBP: Abnormally High: number analyzed (Participants) | 49 | 48 | 48 | 33 | 34 | 31
  SBP: Abnormally High | 42.9 | 45.8 | 35.4 | 18.2 | 17.6 | 12.9
  Diastolic Blood Pressure (DBP): Abnormally Low: number analyzed (Participants) | 49 | 48 | 48 | 33 | 34 | 31
  Diastolic Blood Pressure (DBP): Abnormally Low | 8.2 | 18.8 | 25.0 | 15.2 | 2.9 | 0
  DBP: Abnormally High: number analyzed (Participants) | 49 | 48 | 48 | 33 | 34 | 31
  DBP: Abnormally High | 28.6 | 35.4 | 27.1 | 9.1 | 17.6 | 6.5
  Pulse rate: Abnormally High: number analyzed (Participants) | 49 | 48 | 48 | 33 | 34 | 31
  Pulse rate: Abnormally High | 30.6 | 27.1 | 27.1 | 12.1 | 20.6 | 16.1
  Pulse rate: Abnormally Low: number analyzed (Participants) | 49 | 48 | 48 | 33 | 34 | 31
  Pulse rate: Abnormally Low | 0.0 | 2.1 | 0 | 6.1 | 5.9 | 16.1
  Respiratory rate: Abnormally High: number analyzed (Participants) | 49 | 48 | 48 | 34 | 34 | 31
  Respiratory rate: Abnormally High | 4.1 | 12.5 | 18.8 | 3.1 | 2.9 | 6.5
  Respiratory rate: Abnormally Low: number analyzed (Participants) | 49 | 48 | 48 | 34 | 34 | 31
  Respiratory rate: Abnormally Low | 12.2 | 10.4 | 0.0 | 0 | 0 | 0
  Temperature: Abnormally High | 30.6 | 41.7 | 22.9 | 50.0 | 52.9 | 54.8
  Oxygen saturation: Abnormally Low: number analyzed (Participants) | 50 | 49 | 48 | 32 | 32 | 30
  Oxygen saturation: Abnormally Low | 8.2 | 12.5 | 6.3 | 3.1 | 9.4 | 0

43. Secondary Outcome: Cohort 1: Area Under the Plasma Concentration-Time Curve From Timepoint 0 Hours Until 24 Hours Post Dose (AUC[0-24 Hours])
Description: AUC (0-24) is defined as area under the plasma concentration-time curve from timepoint 0 hours until 24 hours post dose estimated by population PK model.
Time Frame: 0 to 24 hours post dose on Days 1 and 7
Population: PK analysis set included all participants from Cohort-1 who received JNJ-53718678 and for whom at least one PK concentration was reported. Here, 'n' (number analyzed) represents number of participants who were evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: Nanograms*hours per milliliter (ng*h/mL)
Arm/Group | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 30 | 32
Nanograms*hours per milliliter (ng*h/mL)
  >=28 days to <3 months: Day 1: number analyzed (Participants) | 6 | 7
  >=28 days to <3 months: Day 1 | 6690 (1950) | 20600 (3990)
  >=28 days to<3 months: Day 7: number analyzed (Participants) | 6 | 7
  >=28 days to<3 months: Day 7 | 11400 (3930) | 36000 (8140)
  >=3 months to <6 months: Day 1: number analyzed (Participants) | 6 | 4
  >=3 months to <6 months: Day 1 | 5340 (2670) | 23600 (12500)
  >=3 months to <6 months: Day 7: number analyzed (Participants) | 6 | 4
  >=3 months to <6 months: Day 7 | 7370 (4270) | 35000 (20100)
  >=6 months to <=3 years: Day 1: number analyzed (Participants) | 11 | 17
  >=6 months to <=3 years: Day 1 | 6910 (2900) | 25000 (11600)
  >=6 months to <=3 years: Day 7: number analyzed (Participants) | 11 | 17
  >=6 months to <=3 years: Day 7 | 8160 (3950) | 31000 (16300)

44. Secondary Outcome: Cohort 1: Maximum Plasma Concentration (Cmax) of JNJ-53718678
Description: Cmax is the maximum plasma concentration of JNJ-53718678 estimated by population PK model.
Time Frame: Days 1 and 7
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 30 | 32
Nanograms per milliliter (ng/mL)
  >=28 days to <3 months: Day 1: number analyzed (Participants) | 6 | 7
  >=28 days to <3 months: Day 1 | 531 (193) | 1590 (345)
  >=28 days to <3 months: Day 7: number analyzed (Participants) | 6 | 7
  >=28 days to <3 months: Day 7 | 843 (255) | 2550 (550)
  >=3 months to <6 months: Day 1: number analyzed (Participants) | 6 | 4
  >=3 months to <6 months: Day 1 | 497 (256) | 2070 (1200)
  >=3 months to <6 months: Day 7: number analyzed (Participants) | 6 | 4
  >=3 months to <6 months: Day 7 | 691 (306) | 2920 (1500)
  >=6 months to <=3 years: Day 1: number analyzed (Participants) | 12 | 18
  >=6 months to <=3 years: Day 1 | 846 (268) | 2720 (1040)
  >=6 months to <=3 years: Day 7: number analyzed (Participants) | 11 | 17
  >=6 months to <=3 years: Day 7 | 1030 (310) | 3560 (1330)

45. Secondary Outcome: Cohort 1: Trough Plasma Concentration (Ctrough) of JNJ-53718678
Description: Ctrough is the trough plasma concentration of JNJ-53718678 estimated by population PK model.
Time Frame: Days 1 and 7
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose
Number analyzed (Participants) | 30 | 32
ng/mL
  >=28 days to <3 months: Day 1: number analyzed (Participants) | 6 | 7
  >=28 days to <3 months: Day 1 | 64 (31.3) | 167 (147)
  >=28 days to <3 months: Day 7: number analyzed (Participants) | 6 | 7
  >=28 days to <3 months: Day 7 | 267 (111) | 885 (239)
  >=3 months to <6 months: Day 1: number analyzed (Participants) | 6 | 4
  >=3 months to <6 months: Day 1 | 55.5 (33.5) | 204 (58.5)
  >=3 months to <6 months: Day 7: number analyzed (Participants) | 6 | 4
  >=3 months to <6 months: Day 7 | 126 (103) | 702 (487)
  >=6 months to <=3 years: Day 1: number analyzed (Participants) | 11 | 17
  >=6 months to <=3 years: Day 1 | 59.9 (43) | 227 (149)
  >=6 months to <=3 years: Day 7: number analyzed (Participants) | 11 | 17
  >=6 months to <=3 years: Day 7 | 89 (73.6) | 386 (331)

46. Secondary Outcome: Cohort 2: Plasma Concentration of JNJ-53718678
Description: Plasma concentration of JNJ-53718678 was measured for Cohort-2. As per planned analysis in the protocol, PK sampling was performed on either Day 3 or Day 5 for participants receiving twice daily dosing, resulting in one combined timepoint of Day 3 or Day 5. Hence, the data collected on either Day 3 or Day 5 was pooled and is reported here collectively.
Time Frame: Once daily dosing: Day 3 and Day 8 pre- or post-dose. Twice daily dosing: Day 1 at least 1 hour post-dose, and Days 3 or 5 (combined in one timepoint) at least 4 hours after morning dose but prior to evening dose
Population: PK analysis set included all participants from Cohort-2 who received JNJ-53718678 and for whom at least one PK concentration was reported. Here, 'n' (number analyzed) represents number of participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 33 | 30
ng/mL
  Day 3 (Once daily): number analyzed (Participants) | 22 | 21
  Day 3 (Once daily) | 392.97 (638.253) | 931.66 (1757.958)
  Day 8 (Once daily): number analyzed (Participants) | 22 | 20
  Day 8 (Once daily) | 59.05 (84.552) | 364.73 (951.896)
  Day 1 (Twice daily): number analyzed (Participants) | 10 | 7
  Day 1 (Twice daily) | 394.58 (297.539) | 1539.43 (602.591)
  Day 3 or Day 5 (Twice daily): number analyzed (Participants) | 10 | 9
  Day 3 or Day 5 (Twice daily) | 441.13 (305.450) | 1050.44 (663.166)

47. Secondary Outcome: Percentage of Participants With Medical Resource Utilization (MRU)
Description: Percentage of participants with MRU (any medical care encounters) was reported.
Time Frame: Up to Day 28
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 47 | 47 | 44 | 32 | 33 | 28
Percentage of Participants | 100.0 | 100.0 | 100.0 | 9.4 | 15.2 | 25.0

48. Secondary Outcome: Percentage of Participants With Acceptability and Palatability of the JNJ-53718678 Formulation as Assessed by Parent(s)/Caregiver(s)
Description: Percentage of participants with acceptability and palatability of the JNJ-53718678 formulation was assessed through a questionnaire asking about the child's reaction when given the medicine, completed by parent(s)/caregiver(s) after last dosing that categorized as 1) child took medicine easily, 2) disgusted expressions after tasting medicine, 3) cried after tasting medicine, 4) would not open mouth or turned head away to avoid medicine, 5) spit out or coughed out medicine, 6) gagged, and 7) vomited (within 2 minutes of swallowing medicine). Below results are based on response to "child took medicine easily".
Time Frame: Day 8
Population: as for outcome 10
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 34 | 32 | 37 | 24 | 21 | 21
Percentage of Participants | 67.6 | 84.4 | 73.0 | 70.8 | 90.5 | 85.7

49. Secondary Outcome: Number of Participants With Emerging Variations in the Viral Genome Potentially Associated With Resistance to JNJ-53718678
Description: Number of participants with emerging variations in the viral genome potentially associated with resistance to JNJ-53718678 was reported. Number of participants with F gene sequencing data available and with emerging genetic variations post-baseline as compared to baseline, considering 24 RSV F protein positions of interest (positions 127, 137, 138, 140, 141, 143, 144, 323, 338, 339, 392, 394, 396, 397, 398, 399, 400, 401, 474, 486, 487, 488, 489, and 517) was reported.
Time Frame: Up to Day 21
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
Number analyzed (Participants) | 44 | 43 | 40 | 32 | 29 | 28
Participants | 0 | 0 | 2 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to Day 28
Description: The Safety analysis set included all participants who received at least 1 dose of study agent, and were analyzed as treated, regardless of the randomized treatment group assigned.
Arm/Group | Cohort 1: Placebo | Cohort 1: JNJ-53718678 Low Dose | Cohort 1: JNJ-53718678 High Dose | Cohort 2: Placebo | Cohort 2: JNJ-53718678 Low Dose | Cohort 2: JNJ-53718678 High Dose
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49 | 0/48 | 0/34 | 0/34 | 0/31
Serious Adverse Events (participants affected / at risk) | 4/50 | 5/49 | 2/48 | 2/34 | 2/34 | 3/31
Other Adverse Events (participants affected / at risk) | 28/50 | 29/49 | 30/48 | 14/34 | 20/34 | 13/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Placebo (N=50) | Cohort 1: JNJ-53718678 Low Dose (N=49) | Cohort 1: JNJ-53718678 High Dose (N=48) | Cohort 2: Placebo (N=34) | Cohort 2: JNJ-53718678 Low Dose (N=34) | Cohort 2: JNJ-53718678 High Dose (N=31)
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Coronavirus Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Feeding Disorder (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Placebo (N=50) | Cohort 1: JNJ-53718678 Low Dose (N=49) | Cohort 1: JNJ-53718678 High Dose (N=48) | Cohort 2: Placebo (N=34) | Cohort 2: JNJ-53718678 Low Dose (N=34) | Cohort 2: JNJ-53718678 High Dose (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 2 | 2 | 3 | 0 | 2 | 0
Eye Discharge (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anal Erythema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anorectal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 5 | 5 | 3 | 4
Faeces Soft (Gastrointestinal disorders) | 3 | 0 | 2 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Noninfective Gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Post-Tussive Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 3 | 4 | 1 | 0
Face Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 3 | 3 | 0 | 1 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Candida Nappy Rash (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Exanthema Subitum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fungal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0
Hand-Foot-And-Mouth Disease (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lower Respiratory Tract Infection Bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 6 | 0 | 2 | 1
Oral Candidiasis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0
Otitis Media (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1
Otitis Media Acute (Infections and infestations) | 1 | 2 | 1 | 1 | 0 | 1
Parainfluenzae Virus Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 1
Pneumonia Bacterial (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Rhinovirus Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 3 | 1 | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral Rash (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Arthropod Sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Radial Head Dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Skin Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood Potassium Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Platelet Count Increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Transaminases Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Metabolic Alkalosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Zinc Deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchial Secretion Retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Depth Increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 0 | 2 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperaemia (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT03656510/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT03656510/SAP_001.pdf